Protocol Number: KD025-108

<u>Document Title:</u> An Open-label, Two-part Study Designed to Assess the Absolute Bioavailability of KD025 and to Determine the Mass Balance Recovery, Metabolite Profile and Identification of Metabolite Structures for [14C]-KD025 in Healthy Male Subjects

Statistical Analysis Plan: Version 1.0

Date of Document: 20 May 2019

NCT Number: NCT03907540



# REPORTING AND ANALYSIS PLAN

An open-label, two-part study designed to assess the absolute bioavailability of KD025 and to determine the mass balance recovery, metabolite profile and identification of metabolite structures for [14C]-KD025 in healthy male subjects

**Quotient Study Number:** 

QSC200323

**Sponsor Study Number:** 

KD025-108

Sponsor:

Kadmon Corporation LLC

450 East 29th Street

New York NY 10016

Date of RAP:

20 May 2019

Status of RAP:

Final V1.0

**Document Version History** 

| Version<br>Number | Reason for Update | Updated By: | Date |
|-------------------|---------------------|---------------|-------------|
| V1.0 | Finalisation of RAP | Carla Mariner | 20 May 2019 |

#### SPONSOR/QUOTIENT SCIENCES CONFIDENTIAL

This Reporting and Analysis Plan may not be reproduced or communicated to a third party without the written permission of Kadmon Corporation LLC.

| SpansonQuotient Sciences Confident | isi |
|--------------------------------------------------|------------------------|
| Author | |
| Mart | 20 May 2019 |
| Carle Manifer<br>Lead Statistician (Quotient) | Date |
| Approvers | |
| Ann Davidson | 30May 19. |
| Lead Statistical Programmer (Quotient) | pare |
| dilan | al Hoy 2019 |
| Hazel Ross<br>Lead Pharmacokineticlet (Quotient) | Date U |
| CRII | Date Date |
| Claire Pair Lead Medical Writer (Quotient) , | Date |
| Stuart Wood | 28 Way 2019 |
| Metabolism Lead (Phyrmaron) | Date. |
| Naulsudi | 20MAY 2017 |
| Nand Singh Principal Investigator (Quotient) | DME |
| Olivier Schueller | 20-1-4-1-2-019<br>Date |
| Chemical Development (Kadmon Corporation LLC) | Strangers and |
| Senjay Aggaretal | 20-MAY-1019 |
| Clinical Development (Kadmon Comoration Lt C) | Date ' |

# **Table of Contents**

1

| 1 | Table | of Contents | 3 |
|---|---------|----------------------------------------------------------|----|
| 2 | List of | Abbreviations | 6 |
| 3 | Introdu | uction | 9 |
| | 3.1 | Responsibilities | 0 |
| | 3.2 | Definitions | |
| | 3.2.1 | Subjects Definitions | |
| | 3.2.2 | Definition of Treatments | |
| | 3.2.3 | Definition of Visits | |
| 4 | Object | ives | 10 |
| | 4.1 | Primary Objective | 10 |
| | 4.2 | Secondary Objectives | 10 |
| | 4.3 | Study Endpoints | |
| | 4.3.1 | Primary Endpoints | |
| | 4.3.2 | Secondary Endpoints | 11 |
| 5 | Study l | Design | 11 |
| | 5.1 | Brief Description | |
| | 5.1.1 | Study Plan Part 1 | |
| | 5.1.2 | Study Plan Part 2 | |
| | 5.2 | Study Sample Size | |
| | 5.3 | Subject Numbers (including Replacement Subjects) | |
| | 5.4 | Blinding Issues | 13 |
| 6 | Popula | ations for Analysis | 14 |
| | 6.1 | Safety Population | |
| | 6.2 | Pharmacokinetic Population | |
| | 6.3 | Mass Balance Population | 14 |
| 7 | Subjec | t Disposition, Demographics and Baseline Characteristics | 15 |
| | 7.1 | Screening Failures | |
| | 7.2 | Subject Disposition and Withdrawals | |
| | 7.3 | Analysis Populations | |
| | 7.4 | Analysis Datasets | |
| | 7.5 | Demographic Characteristics and Lifestyle Details | |
| | 7.6 | Medical/Surgical History | 16 |
| | 7.7 | Prior and Concomitant Medication | |
| | 7.8 | Other Baseline Characteristics | 17 |
| 8 | Efficac | у | 17 |
| 9 | Pharma | acokinetics and Mass Balance | 17 |
| | 9.1 | Pharmacokinetic Parameter Estimation | |
| | 9.1.1 | Definition of Pharmacokinetic Parameters | |
| | 9.1.2 | Rules for Pharmacokinetic Parameter Estimation | 18 |

| | 9.2 | Pharmacokinetic Parameter Reporting Specifications | 20 |
|---|---|---|---|
| | 9.2.1 | Bioanalytical and Pharmacokinetic Summary Tables | 21 |
| | 9.2.2 | Bioanalytical and Pharmacokinetic Figures | |
| | 9.2.3 | Bioanalytical and Pharmacokinetic Listings | |
| | 9.2.4 | Statistical Analysis of Pharmacokinetic Parameters | |
| | 9.3 | Mass Balance Parameter Estimation | |
| | 9.3.1 | Definition of Mass Balance Parameters | |
| | 9.3.2 | Rules for Mass Balance Parameter Estimation | |
| | 9.4 | Mass Balance Reporting Specifications | |
| | 9.4.1 | Mass Balance Summary Tables | |
| | 9.4.1 | Mass Balance Figures | |
| | 9.4.3<br>9.4.4 | Mass Balance Listings Statistical Analysis of Mass Balance Parameters | |
| 10 | | Assessments | |
| | • | | |
| | 10.1 | Extent of Exposure and Treatment Compliance | |
| | 10.2 | Meal Details | |
| | 10.3 | Adverse Events | |
| | 10.3.1 | Summary Tables for Adverse Events | 29 |
| | 10.3.2 | Listings for Adverse Events | 31 |
| | 10.4 | Laboratory Evaluations | 31 |
| | 10.4.1 | Summary Tables for Laboratory Evaluations | 31 |
| | 10.4.2 | Listings for Laboratory Evaluations | |
| | 10.5 | Vital Signs | |
| | 10.5.1 | Summary Tables for Vital Signs | |
| | 10.5.2 | Listings for Vital Signs | |
| | 10.6 | ECGs | |
| | 10.6.1 | Summary Tables for ECGs | |
| | 10.6.1 | Listings for ECGs | |
| | 10.0.2 | | |
| | | Body Weight | |
| | 10.8 | Physical Examination | 34 |
| 11 | Interim | Statistical Analyses | 34 |
| 12 | Change | es in the Conduct of the Study or Planned Analysis | 34 |
| | 12.1 | Changes in the Conduct of the Study | 34 |
| | 12.2 | Changes to the Planned Analyses | 34 |
| | 12.3 | Any Other Relevant Changes | |
| 13 | Overall | Considerations | 34 |
| | 13.1 | Statistical Programming and Analysis | 34 |
| | 13.2 | Quality Control of Summary Tables, Figures and Listings | |
| | 13.2.1 | Quality Control - Summary Tables | |
| | 13.2.2 | Quality Control - Figures | |
| | 13.2.3 | Quality Control - Data Listings | |
| 14 | SAS Da | ata Transfer | 37 |
| 15 | Prograi | mming Conventions | 37 |
| 16 | • | · · | |
| 10 | Keierei | nce List | <i>31</i> |

| 17 | Index of Tables | . 38 |
|--------|-------------------------------|------|
| 18 | Index of Figures | . 44 |
| 19 | Index of Listings | .49 |
| 20 | Mock Tables | . 55 |
| Append | ix 1: Part 1 Study Flow Chart | . 78 |
| Append | ix 2: Part 2 Study Flow Chart | 81 |

## 2 List of Abbreviations

<sup>14</sup>C carbon-14

ADaM analysis data model

ADME absorption, distribution, metabolism, excretion

ADR adverse drug reaction

AE adverse event

ATC anatomical therapeutic chemical

BLQ below the limit of quantification

BMI body mass index

BP blood pressure

CDISC Clinical Data Interchange Standards Consortium

CHMP Committee for Medicinal Products for Human Use

CSR clinical study report

CV% coefficient of variation

D 'substantial' decrease from baseline for vital signs parameters

DP decimal place

ECG electrocardiogram

F absolute bioavailability

h hour

H flag used for value that is above normal reference range

HR heart rate

'substantial' increase from baseline for vital signs parameters /

l

increase in QTcF interval from baseline

ICH International Council on Harmonisation

IMP investigational medicinal product

IV intravenous

L flag used for value that is below normal reference range

LLOQ lower limit of quantification

LOCF last observation carried forward

Max maximum

MedDRA Medical Dictionary for Regulatory Activities

Min minimum

n number of subjects with an observation

N number of subjects in the dataset

NA not applicable

NC not calculated

NMT not more than

NR no result/not reportable

NS no sample

PI principal investigator

PK pharmacokinetic

PT preferred term

QC quality control

QTcF QT interval corrected for heart rate using Fridericia's correction

RAP reporting analysis plan

SAE serious adverse event

SD standard deviation

SDTM study data tabulation model

SF significant figure

SI substantial increase in QTcF interval from baseline

SOC system organ class

SOP standard operating procedure

TEAE treatment-emergent adverse events

TFL tables, figures and listings

# WHO World Health Organisation Abbreviations used for pharmacokinetic and mass balance parameters and flags are defined in Section 9.

**Sponsor/Quotient Sciences Confidential** 

#### 3 Introduction

This document details the following for Quotient Sciences (Quotient) Study QSC200323 (KD025-108):

- criteria to be used for the definition of the analysis populations relating to safety, pharmacokinetic (PK) and mass balance data
- · handling of missing data
- proposed tables, figures and listings (TFLs) for demographic, dosing, PK, mass balance and safety data
- methods for PK parameter estimation

This document has been compiled according to the Quotient standard operating procedure (SOP) "Production of Reporting and Analysis Plans" and has been written based on information contained in the final study protocol, Version 1.0 dated 17 Jan 2019 and non-substantial amendment NSA01 dated 18 Apr 2019.

#### 3.1 Responsibilities

The Data Sciences Department at Quotient will be responsible for the production of the following items using Quotient SOPs: Clinical Data Interchange Standards Consortium (CDISC) study data tabulation model (SDTM) and analysis data model (ADaM) datasets, PK parameter estimation and output, mass balance parameter estimation and output, and safety output; including all summary TFLs; and the clinical study report (CSR).

Quotient will provide two sets of TFLs during the study:

- post database lock TFLs (draft) for Kadmon Corporation LLC (Kadmon) review, and
- post-review TFLs (final) for inclusion into the CSR

Quotient will be responsible for the quality control (QC) of all deliverables prior to the client review (Section 13.2).

Metabolite profiling and structural identification will be the responsibility of Pharmaron, and will be the subject of a separate Analytical Work Plan. These aspects will be reported separately from the CSR as a standalone document.

#### 3.2 Definitions

#### 3.2.1 Subjects Definitions

During the clinical phase of the study, an evaluable subject is defined:

- for Part 1, as a subject who has sufficient data for evaluation of the primary bioavailability objective of the study
- for Part 2, as a subject who has provided biological samples for up to 168 h after drug administration or has demonstrated >90% mass balance recovery, or has <1% of the administered dose eliminated in excreta for two consecutive days, whichever is the sooner

These definitions of an evaluable subject will not be used during the reporting phase including the identification of analysis populations and datasets.

All enrolled subjects are defined as those subjects who signed the informed consent, qualified per the inclusion/exclusion criteria and were allocated a subject number.

#### 3.2.2 Definition of Treatments

Throughout the reporting of the study, treatments will be reported as detailed in Table 1 below:

**Table 1 Study Treatments** 

| Study<br>Part | Treatment | Investigational Medicinal Product | Label used for Reporting Purposes in Tables Figures and Listings |
|---|---|---|---|
| 1 | Α | KD025 Tablet, 200 mg | 200 mg KD025 Oral Tablet |
| 1 | В | [14C]-KD025 solution for infusion, 20 µg/mL (100 µg in 5 mL) | 100 µg [14C]-KD025 IV Infusion |
| 2 | С | [14C]-KD025 capsule, 200 mg | 200 mg [14C]-KD025 Oral Capsule |

#### 3.2.3 Definition of Visits

For clinical data, visits will be referred to as Day throughout this document and will be referred to as Screening, and

- for Part 1: Day -1 (Admission) and Day 1 through to Day 3 (Discharge)
- for Part 2: Day -1 (Admission) and Day 1 through to Day 15 with discharge planned to occur on Day 8 and a follow-up phone call 5 to 7 days after discharge or after the end of the last collection period

Time points within these days are detailed in the schedule of assessments in Appendix 1 for Part 1 and in Appendix 2 for Part 2. For Part 1, PK data of Treatment B will be reported relative to the start of infusion. For all other PK data, time points will be presented relative to the administration time of Treatment A and C, respectively.

Baseline is defined as nominally the last measurement recorded prior to the first dose of investigational medicinal product (IMP) in each study part.

# 4 Objectives

#### 4.1 Primary Objective

The primary objectives of this study are:

- to determine the absolute oral bioavailability of KD025 (Part 1)
- to determine the mass balance recovery after a single oral dose of [14C]-KD025 (Part 2)
- to provide plasma, urine and faecal samples for metabolite profiling and structural identification (Part 2)

#### 4.2 Secondary Objectives

The secondary objectives of this study are:

- to obtain information regarding the oral PK of total radioactivity, KD025 and its metabolites KD025m1 and KD025m2, in plasma
- to obtain information regarding the intravenous (IV) PK of [14C]-KD025 in plasma (Part 1)
- to determine the routes and rates of elimination of [14C]-KD025 and associated total radioactivity (Part 2)
- to evaluate the extent of distribution of total radioactivity into blood cells (Part 2)
- to assess the qualitative and quantitative metabolic profile of [¹⁴C]-KD025 and carry out the structural elucidation of the main metabolites in plasma (accounting for ≥ 10% of circulating total radioactivity) and in urine and faecal samples (accounting for ≥ 10% of administered dose; Part 2)

to provide additional safety and tolerability information for KD025

#### 4.3 Study Endpoints

#### 4.3.1 Primary Endpoints

- absolute bioavailability (F) of KD025
- mass balance recovery of total radioactivity in all excreta (urine and faeces): Ae, %Ae, Cum Ae and Cum %Ae
- collection of plasma, urine and faeces for metabolite profiling and structural identification

#### 4.3.2 Secondary Endpoints

- assessment of oral PK of KD025, KD025m1 and KD025m2 and total radioactivity by calculation of: Tlag, Tmax, Cmax, AUC(0-last), AUC(0-inf), AUC%extrap, lambda-z, T1/2, CL/F (KD025 only), Vz/F (KD025 only) and MRT
- assessment of IV PK of [<sup>14</sup>C]-KD025 by calculation of: Tmax, Cmax, AUC(0-last), AUC(0-inf), AUC%extrap, lambda-z, T1/2, CL, Vz, Vss and MRT
- determination of routes and rates of elimination of <sup>14</sup>C- by metabolite profiling and structural identification in plasma, urine and faeces
- evaluation of whole blood:plasma concentration ratios for total radioactivity
- amount and structure of metabolites in plasma (accounting for ≥ 10% of circulating total radioactivity), urine and faeces (accounting for ≥ 10% of administered dose).
- to provide additional safety and tolerability information for KD025 by assessing: adverse events (AEs), vital signs, electrocardiograms (ECGs), physical examinations and laboratory safety tests

# 5 Study Design

#### 5.1 Brief Description

This is a single centre, non-randomised, open-label, two-part study in 6 healthy male subjects. Subjects must have participated in Part 1 in order to be eligible for Part 2. An overview of the study is presented in Figure 1 and assessment time points are detailed in Appendix 1 for Part 1 and in Appendix 2 for Part 2.

#### 5.1.1 Study Plan Part 1

Part 1 is an open-label, non-randomised single oral dose (tablet) followed by an IV microtracer assessment.

On Day 1, subjects will receive a single dose of KD025 (Treatment A) 30 min after the start of a standard breakfast. Subjects will then receive an IV dose of [14C]-KD025 (100 µg, a 'microdose') containing not more than (NMT) 37 kBq (1000 nCi) [14C], as a 15 min IV infusion (Treatment B), starting 1.75 h after the oral dose administration (Treatment A) ie, starting 15 min before the expected Tmax (2 h) for the oral dose. Subjects will remain resident in the clinic until up to 48 h post-oral dose (ie up to Day 3).

#### 5.1.2 Study Plan Part 2

Part 2 is an open-label, non-randomised absorption, distribution, metabolism, excretion (ADME) assessment.

Following a minimum washout period of 7 days, subjects who participated in Part 1 of the study will be admitted to the clinical unit for participation in Part 2 of the study (on Day -1). On the morning of Day 1, each subject will receive a single oral administration of 200 mg [ $^{14}$ C]-KD025 capsule containing (NMT 9.8 MBq) (215  $\mu$ Ci) [ $^{14}$ C] (Treatment C) 30 min after the start of a standard breakfast.

Subjects will remain resident in the clinic until up to 168 h after dosing (up to Day 8). It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90% or if <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 h periods. This may result in the subjects being discharged as a group prior to completion of the planned residency period. Once the discharge criteria or the planned residency period has been achieved, the subjects will undergo discharge assessments and collection of all samples (blood, urine and faeces) will be stopped.

If mass balance criteria have not been met by all subjects on Day 8, the residency period for the subjects not achieving the release criteria may be extended up to a maximum of 216 h post-dose (Day 10). During the additional residency period only urine and/or faeces will be collected. If the criterion is still not met by Day 10, or if additional residency is not considered appropriate or necessary, then home collections of urine and/or faeces may be requested at the discretion of the investigator for individual subjects. To ensure ongoing wellbeing of the subjects, a follow-up phone call will take place 5 to 7 days post-discharge from the study or after the end of the last collection period.



Figure 1 Study Sequence

#### 5.2 Study Sample Size

No sample size calculation was performed. For a study of this type, a sample size of 6 subjects, to ensure data in 4 evaluable subjects (as defined in Section 3.2.1) is considered appropriate to meet the objectives of the study.

#### 5.3 Subject Numbers (including Replacement Subjects)

This is an open-label, non-randomised study and therefore a randomisation schedule will not be produced.

Subject numbers will be allocated on the morning of dosing in Part 1 according to the code 001 to 006 using the lowest number available.

No replacement subjects are to be used in this study.

#### 5.4 Blinding Issues

This is an open-label, non-randomised study and therefore blinding is not required.

<sup>&</sup>lt;sup>a</sup> Discharge time relative to oral dose, 48 h post-dose.

<sup>&</sup>lt;sup>b</sup> Subjects who participated in Part 1 will be admitted to the clinical unit on Day -1 of Part 2 after a minimum washout period of 7 days.

c If mass balance criteria have not been met by all subjects on Day 8, the residency period for the subjects not achieving the release criteria may be extended up to a maximum of 216 h post-dose (Day 10). During the additional residency period only urine and/or faeces will be collected. If the criterion is still not met by Day 10, or if additional residency is not considered appropriate or necessary, then home collections of urine and/or faeces may be requested at the discretion of the investigator for individual subjects.

# 6 Populations for Analysis

#### 6.1 Safety Population

The safety population will include all subjects who have received at least 1 dose of IMP via either oral administration or IV administration within the study.

The safety population will be confirmed by Quotient with approval from Kadmon after database lock and will be used for the analysis of demographic and baseline characteristics, and all safety data.

#### 6.2 Pharmacokinetic Population

The PK population will include all subjects who have received at least 1 dose of IMP and who satisfy the following criteria for at least 1 profile in either Part 1 or Part 2:

- no missing samples or invalid post-dose analytical results at critical time points (eg around the Cmax)
- no relevant protocol deviations which may impact the study objectives with respect to the PK endpoints
- no relevant AEs such as vomiting (after oral dosing) or infusion site reaction (after IV dosing) which suggest that the whole dose was not available for absorption/delivery for a particular subject

In the event that quantifiable pre-dose concentrations greater than 5% of Cmax are observed, requirements for further action will be agreed with Kadmon and documented at the same time as the PK population and any corresponding dataset(s).

The PK population will be confirmed by Quotient with approval from Kadmon following derivation of all PK parameter estimates.

If required, a PK analysis dataset or datasets may also be documented by Quotient with approval from Kadmon at the same time as the PK population. The PK analysis dataset(s) will be a subset of the PK population.

All enrolled subjects will be used for the PK data listings and the PK population will be used for the provision of PK tables and figures. The PK analysis dataset(s) may be used instead of the PK population for generation of PK tables and figures or to generate additional PK tables and figures. Where possible, this decision will be documented at the same time as the PK population and PK analysis dataset(s).

#### 6.3 Mass Balance Population

The mass balance population will be defined for Part 2 and will include all subjects who have received 1 dose of IMP in Part 2 and who have evaluable total radioactivity concentration (urinary and/or faecal) data and who have no protocol deviations that may affect the mass balance analysis. Such protocol deviations would include anything that affects the accurate measurement of the amount of urine/faeces collected or any AEs that may affect the mass balance analysis, for example:

- spillage of urine and/or faeces
- · missing collections
- AEs that may affect the mass balance analysis, such as vomiting of the dose

The mass balance population will be confirmed by Quotient with approval from Kadmon once all urinary and faecal data have been received.

If required, a mass balance analysis dataset or datasets may also be documented by Quotient with approval from Kadmon at the same time as the mass balance population. The mass balance analysis dataset(s) will be a subset of the mass balance population.

All enrolled subjects will be used for the mass balance data listings. The mass balance population will be used for the analysis of the mass balance concentration data and the provision of mass balance tables and figures. The mass balance analysis dataset(s) may be used instead of the mass balance population for generation of mass balance tables and figures or to generate additional mass balance tables and figures. Where possible, this decision will be documented at the same time as the mass balance population and mass balance analysis dataset(s).

# 7 Subject Disposition, Demographics and Baseline Characteristics

No formal statistical testing will be performed on subject disposition, or on demographic or baseline data. Summaries of subject disposition and analysis populations will be based on all subjects and summaries of all other data described in this section will be based on the safety population, unless otherwise stated.

#### 7.1 Screening Failures

Data for subjects who have failed screening will be databased but will not be subjected to data cleaning and therefore will not be reported, ie will not be included in the STDM or ADaM datasets, or any of the TFLs or the CSR.

#### 7.2 Subject Disposition and Withdrawals

The number and percentage of subjects enrolled, dosed (in Part 1 and Part 2 separately), completed and discontinued will be presented overall. If any subjects discontinued from the study early then the number of subjects for each reason for discontinuation will be presented overall. However, if none of the subjects discontinued from the study early, then the reasons for discontinuation will not be populated in the summary table.

Subject disposition and withdrawal data will be listed including details of informed consent.

Protocol deviations and any violations of the inclusion/exclusion criteria will also be listed.

#### 7.3 Analysis Populations

A single summary table will be produced detailing the number and percentage of subjects in each population for each study part (for safety and PK populations) and overall (for safety, PK and mass balance populations). The reasons for exclusion from each population will also be included in the summary.

Details of subjects included and excluded in the different analysis populations will be listed.

#### 7.4 Analysis Datasets

If applicable, a summary table per population will be produced detailing the number and percentage of subjects in each analysis dataset for each study part and overall, as required. The table will be based on the relevant population the dataset is a subset of (ie the PK or mass

balance population). The reasons for exclusion from each dataset will also be included in the summary.

Details of subjects included and excluded in the different analysis datasets will be listed.

#### 7.5 Demographic Characteristics and Lifestyle Details

Demographic data (date of birth, ethnicity, race, sex, height [cm], weight [kg] and body mass index [BMI; kg/m²]) will be recorded at screening. Note: Weight is also recorded at admission to Part 2, this data will be listed but not summarised (see Section 10.7). Age will be calculated using the following formula:

and will be rounded down to the nearest year (using the SAS Software floor function). If any subjects are enrolled but not dosed and had other assessments recorded, age will be calculated using the date of informed consent.

Summary statistics (number of subjects with an observation [n], mean, standard deviation [SD], median, minimum and maximum) will be presented overall for age at first dose and for height, weight and BMI at screening. The number and percentage of subjects will be presented overall for race, ethnicity and sex. The denominator for the percentage is all subjects in the safety population. If any values are missing, a "missing" row will be presented on the table.

Lifestyle details (ie smoking history [does the subject smoke, use e-cigarettes or use nicotine replacement products?] and alcohol consumption) will be summarised overall as a categorical variable.

Demographic and lifestyle data for all subjects will be listed.

#### 7.6 Medical/Surgical History

Medical/surgical history will be recorded for each subject at the screening visit and updated at admission to each study part. All medical/surgical history data will be listed by subject.

#### 7.7 Prior and Concomitant Medication

Medications (drug name) will be coded using the World Health Organisation (WHO) Drug Dictionary Global Drug Reference (2019 Q1 version or more recent version) using the following Anatomical Therapeutic Chemical (ATC) classification codes:

- product name
- preferred name
- drug code
- therapeutic subgroup (ATC 2nd level name and code)
- chemical subgroup (ATC 4th level name and code)

Prior medications are defined as medications that starts and stop prior to the first dose of IMP. All other medications will be defined as concomitant medications including those that start prior to the first dose of IMP and continue thereafter. Any medications with an unknown start or stop date will be assumed to be concomitant medications unless a partial start or stop date indicates otherwise.

All medications, including coded terms, will be listed. One combined data listing of prior and concomitant medications will be provided. All prior medications as defined above will be flagged with a "#" symbol. Within this flagged group, medications that started after screening and stopped before dosing of IMP will also be flagged using a "\*" symbol.

#### 7.8 Other Baseline Characteristics

All other baseline characteristics, as listed below, at screening and on admission (unless otherwise stated) for each part (as appropriate) will be listed by subject for all subjects:

- carbon monoxide breath test
- urine drug screen
- · alcohol breath test
- virology (screening only)
- creatinine clearance (screening only)

# 8 Efficacy

Not applicable.

## 9 Pharmacokinetics and Mass Balance

#### 9.1 Pharmacokinetic Parameter Estimation

The PK parameters for [14C]-KD025 (Part 1 IV dose), KD025 (Oral dose in Part 1 and Part 2), KD025m1 (Part 2) and KD025m2 (Part 2) and total radioactivity (Part 2) in plasma will be estimated where possible and appropriate for each subject using Phoenix WinNonlin software (v8.0 or a more recent version, Certara USA, Inc., USA).

#### 9.1.1 Definition of Pharmacokinetic Parameters

Plasma PK parameter definitions and reporting specifications are provided in Table 2.

Table 2 Plasma Pharmacokinetic Parameters and Reporting Specifications

| Parameter | Definition | Unit | DP or<br>SF | No. of DP/SF | Study Part |
|---|---|---|---|---|---|
| Tlag | Time prior to the first measurable<br>(non-zero) concentration (oral<br>administration only) | h | DP | 2 | 1+2 |
| Tmax | Time of maximum observed concentration | h. | DP | 2 | 1+2 |
| Cmax | Maximum observed concentration | mass<br>unit/mL | SF | 3 | 1+2 |
| AUC(0-last) | Area under the curve from 0 time to the last measurable concentration | mass<br>unit.h/mL | SF | 3 | 1+2 |
| AUC(0-inf) | Area under the curve from dosing extrapolated to infinity | mass<br>unit.h/mL | SF | 3 | 1+2 |
| AUCextrap | measurable concentration | | DP | 2 | 1+2 |
| T1/2 | Apparent terminal elimination half-<br>life | h | DP | 2 | 1+2 |
| lambda-z | The first order rate constant associated with the terminal (log-linear) portion of the curve | 1/h | DP | 4 | 1+2 |
| CL | Apparent total body clearance after intravenous administration | mL/min | SF | 3 | 1 |

| Parameter | Definition | Unit | DP or<br>SF | No. of DP/SF | Study Part |
|---|---|---|---|---|---|
| CL/F | Apparent total body clearance after extravascular administration, where F (fraction of dose bioavailable) is unknown | mL/min | SF | 3 | 1 + 2ª |
| Vz | Apparent volume of distribution<br>based on the terminal phase after<br>intravenous administration | L | SF | 3 | 1 |
| Vz/F | Apparent volume of distribution based on the terminal phase after extravascular administration, where F (fraction of dose bioavailable) is unknown | L | SF | 3 | 1 + 2ª |
| Vss | Predicted volume of distribution at steady-state after intravenous administration | L | SF | 3 | 1 |
| MRT(0-inf) | Mean residence time extrapolated to infinity (after IV or extravascular administration) | h | DP | 2 | 1+2 |
| F Cmax | Absolute bioavailability of the oral formulation compared to IV based on Cmax | % | DP | 2 | 1+2 |
| F AUC(0-inf) | Absolute bioavailability of the oral formulation compared to IV based on AUC(0-inf) | % | DP | 2 | 1 + 2 |
| Frel Cmax | Relative bioavailability based on<br>Cmax | % | DP | 2 | 1/2ª |
| Frel AUC(0-<br>inf) | Relative bioavailability based on AUC(0-inf) | % | DP | 2 | 1/2ª |
| MPR Cmax | Metabolite to parent ratio based on Cmax | NA | DP | 2 | 2 |
| MPR<br>AUC(0-inf) | Metabolite to parent ratio based on AUC(0-inf) | NA | DP | 2 | 2 |
| lambda-z<br>lower <sup>b</sup> | Lower limit on time for values to be included in the calculation of Lambda-z | h | DP | 2 | 1+2 |
| lambda-z<br>upper <sup>b</sup> | Upper limit on time for values to be included in the calculation of Lambda-z | h | DP | 2 | 1+2 |

DP = decimal places

#### 9.1.2 Rules for Pharmacokinetic Parameter Estimation

For Part 1, PK parameters for Treatment B will be calculated using times relative to the start of infusion. For Treatment A (Part 1) and Treatment C (Part 2), PK parameters will be calculated using times relative to the administration time of Treatment A and C, respectively.

The imputation of non-numerical or negative values reported in the input dataset will be performed as follows:

- pre-dose sample times will be entered as zero
- values that are below the limit of quantification (BLQ) obtained prior to the Cmax will be entered as zero
- values that are BLQ after the Cmax will be treated as missing
- should partial AUCs be required, then values that are BLQ after Cmax may be imputed as zero for these partial areas if lambda-z cannot be determined

SF = significant figures

a = only for KD025

<sup>&</sup>lt;sup>b</sup> = these values should be listed but omitted from the descriptive statistics

NA = not applicable

- values that are quantifiable after at least 2 consecutive BLQ values after Cmax will be treated as missing for the calculation of PK parameters
- values that are reported as "No Result" (NR) or "No Sample" (NS) etc. will be treated as missing

PK parameters will be estimated using standard Phoenix WinNonlin methods, details of which may be found in the documentation accompanying the WinNonlin software package. The following constraints will apply:

| Parameter Estimation | Constraint |
|---|---|
| Sampling times | Actual |
| Trapezoidal method | Linear up / Log down rule |
| Number of points used for lambda-z | At least 3, not including Cmax |
| Minimum requirements for AUC | At least 3 consecutive quantifiable concentrations |
| Dose | Oral: Nominal<br>IV: Actual |
| Rounded dose level | 3 Significant Figures |

Prior to PK parameter estimation the bioanalytical data may be corrected to account for the proportion of administered [¹⁴C] material not measured due to the use of a [¹²C] LC-MS/MS analysis method. Data correction will only be performed if the [¹⁴C]-contribution exceeds 1% of the dose administered. If required, KD025, KD025m1 and KD025m2 bioanalytical data will be multiplied by the determined data correction factor in SAS by the lead statistical programmer (or designee).

Where possible, the terminal elimination rate constant (lambda-z) will be calculated for all subjects. The value of lambda-z will be determined by the slope of the regression line of the natural log transformed concentrations vs time.

The WinNonLin determined choice of data points for determination of lambda-z will be reviewed by the pharmacokineticist who may adjust the selection in order to provide a more appropriate fit. The choice of data points for determination of lambda-z for each profile will be confirmed following a documented peer review.

Absolute Bioavailability of KD025 (F) will be calculated for individual subjects where possible as follows:

$$F = \left\{ \frac{\text{AUC or Cmax (KD025 oral)}}{\text{AUC or Cmax ([14C] - KD025 IV)}} \times \frac{\text{Dose(IV)}}{\text{Dose(oral)}} \right\} \times 100$$

F will be calculated using Cmax and AUC(0-inf). If for any reason the AUC(0-inf) is not calculable (NC), then an alternative or additional AUC such as AUC(0-last) or an AUC over a partial area may be used to calculate F.

The following comparisons will be made:

- absolute bioavailability tablet (Treatment A vs Treatment B)
- absolute bioavailability capsule (Treatment C vs Treatment B)

Non-dose-corrected relative bioavailability (Frel) will be calculated for individual subjects where possible as follows:

$$Frel = \left\{ \frac{AUC \text{ or Cmax (test)}}{AUC \text{ or Cmax (reference)}} \right\} \times 100$$

Frel will be calculated using Cmax and AUC(0-inf). If for any reason the AUC(0-inf) is not calculable then an alternative or additional AUC such as AUC(0-last) over a partial area may be used to calculate Frel.

The following comparisons will be made, where tablet dosing [Treatment A] is considered the reference):

relative bioavailability capsule versus tablet (Treatment C vs Treatment A)

In Part 2, metabolite to parent ratios (MPR) will be calculated as follows using AUC(0-inf) and Cmax. If for any reason the AUC(0-inf) is not calculable then an alternative or additional AUC such as AUC(0-last) may be used:

$$MPR = \frac{AUC \text{ or Cmax (metabolite)}}{AUC \text{ or Cmax (parent)}} \times \frac{MW \text{ (parent)}}{MW \text{ (metabolite)}}$$

Correcting for molecular weight (MW):

- KD025 MW = 452.52 g/mole
- KD025m1 MW= 410.44 g/mole
- KD025m2 MW = 411.42 g/mole

In addition, for Part 2, total radioactivity whole blood to plasma ratios will be determined using SAS by the Lead Statistical Programmer (or designee) at the time points defined in the protocol for whole blood total radioactivity sampling. If the blood and/or plasma concentration values are BLQ (ie less than the lower limit of quantification [LLOQ]) at any given time point, then the ratio will not be calculated.

When converting whole blood collection weights to blood volume (if required) for the calculation of the whole blood to plasma ratios, the following conversion factor will be used:

$$1.06 g of blood = 1 mL of blood$$

This will be calculated in SAS as follows:

Alternatively, where total radioactivity concentrations in whole blood have been provided in mass unit/g units the following conversion will be performed using SAS:

Concentration (mass units/g) \* 1.06 = Concentration (mass units/mL)

#### 9.2 Pharmacokinetic Parameter Reporting Specifications

The following parameters will be reported for each study part and treatment where possible and appropriate, according to the reporting specifications provided in Table 2:

For plasma [14C]-KD025 following IV administration (Part 1)

Tmax, Cmax, AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL, Vz, Vss, MRT(0-inf)

#### For plasma KD025 following oral administration (Part 1)

Tlag, Tmax, Cmax, AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, Vz/F, MRT(0-inf), F Cmax, F AUC(0-inf)

# <u>For plasma Total Radioactivity, KD025, KD025m1 and KD025m2 following oral administration</u> (Part 2)

Tlag, Tmax, Cmax, AUC(0-last), AUC(0-inf), AUCextrap, T1/2, lambda-z, CL/F, Vz/F, MRT(0-inf), F Cmax, F AUC(0-inf), MPR Cmax, MPR AUC(0-inf)

Note: CL/F and Vz/F calculated for KD025 only.

#### For KD025 (Part 1/Part 2) Frel Cmax, Frel AUC(0-inf)

The following flags/footnotes may be applied to the PK parameters:

| Flag | Footnote |
|---|---|
| а | Rsq of regression was <0.9 |
| b | Period used for regression analysis was less than 2-fold the calculated half-life |
| С | Extrapolated portion of AUC(0-inf) >20% |
| d | Insufficient post-Cmax data points for estimation of lambda-z |
| е | Entire profile BLQ, no pharmacokinetic parameters could be calculated |
| f | Quantifiable pre-dose values were observed, however were considered less than 5 % of Cmax |

In the event that the Rsq of regression was <0.9 ('a' flag) or the extrapolated portion of AUC(0-inf) >20% ('c' flag), then lambda-z, AUC(0-inf) and the parameter estimates derived using lambda-z and/or AUC(0-inf), as appropriate, will be deemed unreliable and will be listed but excluded from the summary statistics.

In the event that the period used for regression analysis was less than 2-fold the calculated half-life ('b' flag), parameter estimates derived using lambda-z will be listed, flagged and included in summary statistics.

Additional flags may be applied based on emerging data.

In the event that quantifiable pre-dose values less than 5% of Cmax were observed, all parameter estimates for the profiles affected will be listed, flagged and included in summary statistics.

Note: in the event that quantifiable pre-dose concentrations greater than 5% of Cmax are observed, requirements for further action will be agreed with Kadmon and documented at the same time as the PK population. In this case, an additional flag would be defined.

#### 9.2.1 Bioanalytical and Pharmacokinetic Summary Tables

Summary statistics (ie n, mean, SD, coefficient of variation [CV%], median, minimum, maximum, geometric n, geometric mean, geometric SD and geometric CV%) will be presented for each study part and time point (except pre-dose time points for which geometric summary statistics will not be presented) for the following concentration data where possible:

#### Part 1:

- plasma concentrations of KD025 (following Treatment A)
- plasma concentrations of [14C]-KD025 (following Treatment B)
- Part 2 (following Treatment C):
  - plasma concentrations of KD025, KD025m1 and KD025m2
  - plasma concentrations of total radioactivity
  - whole blood concentrations of total radioactivity
  - whole blood:plasma concentration ratios of total radioactivity

Imputation of non-numerical values reported in the plasma concentration data (ie values that are BLQ) will be entered as zero for the determination of summary statistics with the exception of geometric mean parameters where BLQ values will be imputed as half the LLOQ value. This also applies to any concentrations that are defined as PK parameters.

Summary statistics (ie n, mean, SD, CV%, median, minimum and maximum) will be calculated for all plasma PK parameters by study part and analyte as follows. Geometric n, geometric mean, geometric SD and geometric CV% will be presented for all PK parameters except Tlag and Tmax.

- Part 1:
  - plasma PK parameters of KD025 (following Treatment A)
  - plasma PK parameters of [14C]-KD025 (following Treatment B)
- Part 2 (following Treatment C):
  - plasma PK parameters of KD025, KD025m1 and KD025m2 and total radioactivity
- Part 1/Part 2:
  - Relative Bioavailability of tablet to capsule formulation

Data recorded as not reportable/no result (NR) or no sample (NS) will be handled as missing, ie no assumption will be made about the actual concentration. If applicable, parameters recorded as not calculated (NC) will be handled as missing.

#### 9.2.2 Bioanalytical and Pharmacokinetic Figures

Arithmetic mean concentration vs time curves will be produced on a linear/linear scale and error bars for ± arithmetic SD will be included on the plots.

Geometric mean concentration vs time curves will be produced on a log10/linear scale. Error bars will be included on these plots, where the error bars are (geometric mean ×/÷ geometric SD).

Mean concentration vs time plots (using nominal times) will be produced for on the linear/linear and the log 10/linear scale as follows:

#### Part 1

- KD025 in plasma 1 profile per plot (Treatment A)
- [14C]-KD025 in plasma 1 profile per plot (Treatment B)

#### Part 2

- KD025, KD025m1, KD025m2 and total radioactivity in plasma 4 profiles on the same plot (Treatment C)
- Total radioactivity in plasma and total radioactivity in whole blood 2 profiles on the same plot (Treatment C)

#### Part 1/Part 2

 KD025 in plasma (Treatment A) and KD025 in plasma (Treatment C) – 2 profiles on the same plot

If judged to aid interpretation, the above plots may be produced with or without error bars.

Separate concentration vs time spaghetti plots (using actual sampling time after dosing) will be produced for each study part and analyte (including total radioactivity) for plasma and whole blood with each plot displaying 1 line per profile. These will be produced on the linear/linear and the log 10/linear scale.

Individual concentration vs time plots (using actual sampling times after dosing) will be produced for each individual subject for study part 2 (all analytes, including total radioactivity in plasma and whole blood overlaid).

For all plots on a linear/linear scale, concentration values reported as BLQ will be set to zero. For all plots on a log 10/linear scale, concentration values reported as BLQ will be set to  $\frac{1}{2}$  x LLOQ (except for pre-dose samples on Day 1 which will not be plotted).

Where curves from multiple treatments, analytes or subjects are overlaid on the same plot, symbols will be used to identify different subjects/ treatment regimens and a legend will be included on the plots to define the symbols used.

#### 9.2.3 Bioanalytical and Pharmacokinetic Listings

The sample collection data (eg collection times) for PK samples will be listed. In addition, all concentration data including individual ratios (total radioactivity whole blood:plasma) and PK parameters will be listed on a per subject basis. Any flags used will be given with the appropriate definition.

#### 9.2.4 Statistical Analysis of Pharmacokinetic Parameters

No formal statistical analysis will be performed for the PK data in this study. Descriptive statistics are considered adequate for a study of this type.

#### 9.3 Mass Balance Parameter Estimation

For Part 2, Pharmaron will provide the following concentration and weight data on a per subject basis for each collection interval as specified in the clinical protocol:

- total radioactivity concentration (mass unit equivalents/g) for each of urine and faeces
- weight of urine (g)
- faeces weight (g) ie not faecal homogenate weight

Concentration values will be expressed in terms of mass unit equivalents of the free base form. Quotient Data Sciences will be responsible for the calculation of excretion and recovery of total radioactivity in urine, faeces and urine and faeces combined for inclusion into the CSR. For the purposes of this document, "excretion" will be used when describing the amount of total radioactivity excreted and "recovery" will be used when describing the amount of total radioactivity expressed as a percentage of the radioactive dose administered.

#### 9.3.1 Definition of Mass Balance Parameters

A list of mass balance parameter definitions with reporting specifications are provided in Table 3.

**Table 3 Mass Balance Parameters and Reporting Specifications** 

| Parameter Definition | | Units | DP or SF | No. of<br>DP/SF |
|---|---|---|---|---|
| Ae(urine) | amount of total radioactivity excreted in urine | Mass unit equiv | SF | 3 |
| %Ae(urine) | amount of total radioactivity excreted in urine expressed as a percentage of the radioactive dose administered | % | DP | 2 |
| CumAe(urine) | cumulative amount of total radioactivity excreted in urine | Mass unit equiv | SF | 3 |
| Cum%Ae(urine) cumulative amount of total radioactivity excreted in urine expressed as a percentage of the radioactive dose administered | | % | DP | 2 |
| Ae(faeces) | amount of total radioactivity excreted in faeces | Mass unit equiv | SF | 3 |
| %Ae(faeces) | amount of total radioactivity excreted in faeces expressed as a percentage of the radioactive dose administered | . % | DP | 2 |
| CumAe(faeces) | cumulative amount of total radioactivity excreted in faeces | Mass unit equiv | SF | 3 |
| Cum%Ae(faeces) | cumulative amount of total | | DP | 2 |
| Ae(total) | amount of total radioactivity excreted in urine and faeces combined | Mass unit equiv | SF | 3 |
| %Ae(total) amount of total radioactivity excreted in urine and faeces combined expressed as a percentage of the radioactive dose administered | | % | DP | 2 |
| CumAe(total) | cumulative amount of total<br>radioactivity excreted in urine and<br>faeces combined | Mass unit equiv | SF | 3 |
| Cum%Ae(total) | cumulative amount of total radioactivity excreted in urine and faeces combined expressed as a percentage of the radioactive dose administered | <b>%</b> | DP | 2 |

DP=decimal places

SF=significant figures

Home collections of urine and/or faeces may be requested at the discretion of the investigator for individual subjects. All mass balance parameters will be calculated over all available time points, including home collection, if applicable.

#### 9.3.2 Rules for Mass Balance Parameter Estimation

The following will be calculated for total radioactivity in urine, faeces and urine and faeces combined (ie total) by Quotient Data Sciences (note that the amount excreted in pre-dose samples will not be included in the calculation of the cumulative amount excreted or in the calculation of the cumulative percentage of the radioactive dose excreted):

 the amount excreted in urine, ie Ae(urine), and the amount excreted in faeces, ie Ae(faeces), will be calculated for each collection interval using the following formula (where matrix is either urine or faeces):

• the total amount excreted in urine and faeces combined, ie Ae(total), will be calculated for each collection interval using the following formula:

- the cumulative amount excreted in urine, ie CumAe(urine), and the cumulative amount excreted in faeces, ie CumAe(faeces), will be calculated by the incremental summation of the Ae(<matrix>) across all collection intervals (where matrix is either urine or faeces). The amount excreted in the pre-dose sample should not be included in the calculation of the cumulative amount excreted.
- the cumulative amount excreted in urine and faeces combined, ie CumAe(total), will be calculated across all collection intervals using the following formula:

• the % recovery of the total radioactive dose in urine, ie %Ae(urine), and the % amount of the total radioactive dose excreted in faeces, ie %Ae(faeces), will be calculated for each collection interval using the following formula (where matrix is either urine or faeces):

the % recovery of the total radioactive dose in urine and faeces combined, ie %Ae(total),
 will be calculated for each collection interval using the following formula:

$$%Ae(total) = %Ae(urine) + %Ae(faeces)$$

- the cumulative % amount of the total radioactive dose excreted in urine, ie Cum%Ae(urine), and the cumulative % amount of the total radioactive dose excreted in faeces, ie Cum%Ae(faeces), will be calculated by the incremental summation of the %Ae(<matrix>) across all collection intervals (where matrix is either urine or faeces). The % amount of the total radioactive dose excreted in the pre-dose sample should not be included in the calculation of the cumulative % of dose excreted.
- the cumulative % amount of the total radioactive dose excreted in urine and faeces combined, ie Cum%Ae(total), will be calculated for each collection interval using the following formula:

For urine and faeces, where a subject has failed to void over a particular collection interval the amount excreted (Ae) will be set to zero.

If part of a void over a particular collection interval is missing due to spillage or accidental discarding, the Ae will still be calculated providing other samples have been collected within the interval. Where no other samples are collected within the interval, the data will be set to missing for the purposes of the calculation of Ae, %Ae, CumAe and Cum%Ae. In both scenarios the data will be flagged to highlight a missing void.

Imputation of non-numerical values reported in the urine and faecal dataset (ie concentrations that are BLQ) will be entered as zero for calculation of parameters.

When converting urine collection weights to urine volume (if required), the following conversion factor will be used:

1.02 g of urine = 1 mL of urine

This will be calculated in SAS as follows:

*Urine weight (g) / 1.02 = Urine volume (mL)* 

If total radioactivity concentrations in urine have been provided in mass unit/g units, the following conversion (if required) will be performed using SAS:

Concentration (mass units/g) \* 1.02 = Concentration (mass units/mL)

The radioactivity associated with toilet paper may be determined if considered necessary. The results will be reported for each subject as a single value for the whole collection period and included in the calculation of overall cumulative excretion and recovery parameters.

The following dose levels will be used for mass balance analysis and will be applied with the following constraints:

| Radioactive dose level for mass balance analysis | Actual |
|--------------------------------------------------|-----------------------|
| Rounded dose level | 3 significant figures |

#### 9.4 Mass Balance Reporting Specifications

#### 9.4.1 Mass Balance Summary Tables

Summary statistics (ie n, mean, SD, CV%, median, minimum and maximum) will be presented for amount excreted (Ae) and recovery (%Ae) by collection period for the following:

- urine, ie Ae(urine) and %Ae(urine), for total radioactivity
- faeces, ie Ae(faeces) and %Ae(faeces), for total radioactivity
- urine and faeces combined, ie Ae(total) and %Ae(total), for total radioactivity

In addition, summary statistics (ie n, mean, SD, CV%, median, minimum and maximum) will be presented for cumulative excretion (CumAe) and cumulative recovery (Cum%Ae) by collection period and for the study as a whole for each of the following:

- urine, ie CumAe(urine) and Cum%Ae(urine), for total radioactivity
- faeces, ie CumAe(faeces) and Cum%Ae(faeces), for total radioactivity

urine and faeces combined, ie CumAe(total) and Cum%Ae(total), for total radioactivity

If any subject withdraws prior to the end of a study visit or if subjects have differing collection intervals (eg collection to Day 8 for some subjects and Day 10 for others), then a last observation carried forward (LOCF) approach will also be used whilst calculating cumulative parameters (ie CumAe and Cum%Ae), where the last observed value will be carried forward to the subsequent time point. If this is the case, then 2 tables will be presented. The first table will have the observed values without the use of LOCF so the number of subjects may reduce over time and the second table will have the LOCF values included so that the number of subjects will remain constant over time. Table numbering will be revised as applicable.

#### 9.4.2 Mass Balance Figures

Mass balance figures will be presented for the mass balance population.

Arithmetic mean cumulative excretion (ie CumAe) and cumulative recovery (ie Cum%Ae) vs time curves will be produced on a linear/linear scale and will include ± SD bars. This means there will be 2 plots:

- one plot with CumAe(urine), CumAe(faeces) and CumAe(total) for total radioactivity in plasma overlaid
- a separate plot with Cum%Ae(urine), Cum%Ae(faeces) and Cum%Ae(total) for total radioactivity in plasma overlaid

A legend identifying each profile (ie urine, faeces and total) will be displayed on the mean plots. Figures will be produced using the LOCF imputation strategy (see Section 9.4.1) if summary tables are produced for this method.

#### 9.4.3 Mass Balance Listings

The sample collection data (eg collection intervals) for all urine and faecal samples will be listed. In addition, all total radioactivity concentrations, urine and faecal weights and all mass balance parameters will be listed on a per subject basis.

#### 9.4.4 Statistical Analysis of Mass Balance Parameters

No formal statistical analysis is required for the mass balance data in this study. Descriptive statistics are considered adequate for a study of this type.

# 10 Safety Assessments

The safety population will be used for all safety data summaries.

Separate summary tables and listings will be produced for each study part, unless otherwise specified. Screening data for ECGs and vital signs will be listed only once, under Part 1 listings.

For Part 1, safety data and related summaries will be based on the combination of both regimens associated with the study part, rather than being presented in relation to a specific treatment, unless otherwise specified.

#### 10.1 Extent of Exposure and Treatment Compliance

In Part 1, the dose of Treatment B, including the dose of radioactivity (in kBq), will be summarised (ie, n, mean, SD, median, minimum and maximum). In addition, the number of subjects exposed to Treatment A will also be presented.

In Part 2, the dose of Treatment C, including the dose of radioactivity (in MBq and  $\mu$ Ci), will be summarised (ie, n, mean, SD, median, minimum and maximum).

Dosing details (including the date and time of all doses administered) will be listed for all subjects. Any recorded deviations from the planned dosing regimen will be listed as protocol deviations.

#### 10.2 Meal Details

Meal details as recorded in the database will be listed. Any recorded deviations from the planned meal times will be listed as protocol deviations.

#### 10.3 Adverse Events

Throughout the study, all AEs will be evaluated by the principal investigator (PI) and noted in the AE section of the study database.

For Part 1, AEs will be assigned to the combination of both regimens associated with the study part and not assigned to a specific treatment.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA v22.0), and reported by System Organ Class (SOC) and Preferred Term (PT).

Adverse events will be classified into the following categories:

- pre-dose AEs: AEs recorded at screening or with a start date and time prior to the first dose of IMP
- treatment-emergent adverse events (TEAEs): AEs that commence during/after the first dose of IMP or commence before first dose of IMP (ie a pre-dose AE or existing medical condition) but worsen in intensity during exposure to IMP.

Where the severity of a pre-dose AE intensifies during/after dosing this will be defined as a new AE and classified as a TEAE.

TEAEs will be assigned to the study part in which the AE first occurred. Where the severity of an AE intensifies or symptoms change in a subsequent study part, this will be defined as a new AE and included under the treatment(s) associated with the subsequent study part. Adverse events that occur during the washout period will be assigned to the study part [treatment(s)] the subject received during the period immediately before the washout period.

Adverse events will be classified as "unrelated", "possibly related" and "related" when considering their relationship to IMP. TEAEs classified as "possibly related" and "related" will be defined as adverse drug reactions (ADRs). An ADR is any AE where a causal relationship with the IMP is at least reasonable possibility (ie "possibly related" and "related"). Pre-dose AEs will always have the classification of "unrelated".

Adverse events will be classified as "mild," "moderate" or "severe" when considering their severity.

If the severity or relationship to IMP of a TEAE is missing, the severity/relationship will be tabulated as "missing" in the summary tables.

Where the start date of an AE is missing and the stop date is on or after the day of first dose of IMP or both the start and stop dates are missing then a "worst-case" scenario will be assumed (ie the AE is assumed to have occurred post-dose and is therefore considered

treatment-emergent). If a partial start date/time is available then the event will be considered as treatment-emergent unless the partial information suggests otherwise. The study part to which the AE will be assigned will be programmatically assigned in SAS.

#### 10.3.1 Summary Tables for Adverse Events

All pre-dose AEs (as defined in Section 10.3) will be excluded from the summary tables but will be listed for all subjects.

Descriptive statistical methods will be used to summarise the TEAE data.

The number and percentage of subjects reporting each TEAE will be summarised for both SOC and PT. For summaries by SOC and PT, with the exception of TEAEs by severity and relationship to IMP, the number of subjects and the number of events will be summarised. For summaries by severity and relationship only the number of subjects will be summarised.

For counts of subjects experiencing events the following will apply:

- a subject experiencing TEAEs in more than one body system, within a study part, will be counted once in the total number of subjects with TEAEs in that study part
- a subject with more than 1 TEAE in the same SOC, within a study part, counts only once at the SOC level:
- a subject with more than 1 TEAE in the same PT, within a study part, counts only once at the PT level.

For event counts, all events are included.

When it is necessary to calculate percentages, the denominator will be the total number of subjects in the safety population for that study part and the numerator will be the total number of subjects reporting a TEAE within the relevant category.

Summaries presented for SOC and PT will be presented in descending order of frequency overall (ie most frequently reported SOC in the study part and then by most frequently reported PT in the study part within each SOC).

#### 10.3.1.1 Overall Summary of Adverse Events

The following will be summarised for the safety population by study part:

- number and percentage of subjects reporting at least one TEAE
- number and percentage of subjects reporting ADRs
- number and percentage of subjects reporting severe TEAEs
- number and percentage of subjects reporting serious TEAEs
- number and percentage of subjects reporting TEAEs leading to subject withdrawal
- number and percentage of subjects reporting TEAEs leading to death
- total number of TEAEs
- total number of ADRs
- total number of severe TEAEs
- total number of serious TEAEs
- total number of TEAEs leading to subject withdrawal
- · total number of TEAEs leading to death

# 10.3.1.2 Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

All subjects reporting TEAEs will be summarised by study part. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 TEAE within a study part will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by study part. Counts will be given for number of subjects and number of events. For programming purposes counts of number of subjects will be by maximum severity (ie subjects experiencing more than 1 episode of a TEAE within a study part will be counted only once within each SOC and PT using the most severe episode).

#### 10.3.1.3 Summary of Treatment-Emergent Adverse Events by Severity

All subjects reporting TEAEs will be summarised by severity of TEAE (mild, moderate or severe) and study part. Counts will be given for number of subjects, not number of events. Counts will be given by maximum severity (ie subjects experiencing more than 1 TEAE within a study part will be counted only once using the most severe episode).

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by maximum severity (ie mild, moderate or severe) and study part. Counts will be given for total number of subjects, not for events. Counts by maximum severity will be given (ie subjects experiencing more than 1 TEAE within a study part will be counted only once within each SOC and PT using the most severe episode).

#### 10.3.1.4 Summary of Treatment-Emergent Adverse Events by Relationship to IMP

All subjects reporting TEAEs will be summarised by relationship to IMP (ie unrelated, possibly related and related) and study part. Counts will be given for number of subjects, not number of events. Counts will be given by the closest relationship to IMP (ie subjects experiencing more than 1 TEAE within a study part will be counted only once using the most closely related event).

Additionally, subjects reporting TEAEs will be summarised for SOC and PT by closest relationship to IMP (ie unrelated, possibly related or related) and study part. Counts will be given for total number of subjects, not for events. Counts by closest relationship will be given (ie subjects experiencing more than 1 TEAE within a study part will be counted only once within each SOC and PT using the most closely related event).

#### 10.3.1.5 Summary of Adverse Drug Reactions

All subjects reporting ADRs will be summarised by study part. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 ADR within a study part will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting ADRs will be summarised for SOC and PT by study part. Counts will be given for number of subjects and number of events. For programming purposes counts of number of subjects will be by maximum severity (ie subjects experiencing more than 1 episode of a TEAE within a study part will be counted only once within each SOC and PT using the most severe episode).

#### 10.3.1.6 Summary of Serious Adverse Events

All subjects reporting serious adverse events (SAEs) will be summarised by study part. Counts will be given for number of subjects and number of events. Subjects experiencing more than 1 SAE within a study part will be counted only once for number of subjects but will be counted more than once for number of events.

Additionally, subjects reporting SAEs will be summarised for SOC and PT by study part. Counts will be given for number of subjects and number of events. For programming purposes counts of number of subjects will be by maximum severity (ie subjects experiencing more than 1 episode of a SAE within a study part will be counted only once within each SOC and PT using the most severe episode).

#### 10.3.2 Listings for Adverse Events

All pre-dose AEs (as defined in Section 10.3) will be listed including SOC and PT.

A separate data listing of all TEAEs will be provided for each study part including the SOC and PT. In addition a listing of all SAEs will be provided.

#### 10.4 Laboratory Evaluations

The details of sample collection for laboratory safety analysis are described in the study protocol.

Where a value is provided by the safety laboratory as either above or below the limit of detection this will be set to the limit of detection itself for summary purposes. No imputations will be made in the individual listings.

#### 10.4.1 Summary Tables for Laboratory Evaluations

Haematology and clinical chemistry data will be summarised (n, mean, SD, median, minimum and maximum) for each laboratory parameter at each time point, including changes from baseline (Day 1, Pre-dose for each study part) to Day 3 in Part 1 and Day 8 in Part 2 by study part. Shift tables from baseline to Day 3 in Part 1 and Day 8 in Part 2 by study part (with respect to the number and percentage of subjects with values below, within or above the reference range) will be presented by study part. Percentages will be based on the number of subjects with measurements at baseline and the relevant post-baseline time point.

Reference ranges for each laboratory parameter will be presented for the relevant parameter in each summary table.

#### 10.4.2 Listings for Laboratory Evaluations

The sample collection data (eg collection times) for laboratory analysis and urinalysis data will be listed.

All individual subject data, for planned haematology, clinical chemistry, and urinalysis data including derivations such as change from baseline will be listed. If applicable, data from unscheduled laboratory tests will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics. In these listings, individual data will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively.

Separate listings of all haematology, clinical chemistry and urinalysis values outside their reference ranges by subject will also be provided. References ranges will be supplied by the safety laboratory for haematology and clinical chemistry and per the database for urinalysis (ie a positive or negative result) with the exception of the following reference ranges for urinalysis:

• pH: 5.0 to 9.0

Specific gravity: 1.000 to 1.030

#### 10.5 Vital Signs

The details of measurement of supine vital signs are described in the study protocol.

#### 10.5.1 Summary Tables for Vital Signs

Vital signs data (ie systolic and diastolic blood pressure [BP], heart rate and oral body temperature), including change from baseline (Day 1, Pre-dose for each study part), will be summarised (ie n, mean, SD, median, minimum and maximum) at each post-baseline time point by study part.

In addition, the number of subjects with 'substantial' increases or decreases or no substantial change from baseline in systolic BP ( $>\pm20$  mmHg), diastolic BP ( $>\pm10$  mmHg) and heart rate ( $>\pm15$  bpm) will be summarised.

#### 10.5.2 Listings for Vital Signs

All individual vital signs data (ie systolic and diastolic BP, heart rate and oral body temperature), including derivations such as change from baseline will be listed. Individual data will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively, and subjects with 'substantial' increases or decreases from baseline (as defined in Section 10.5.1) in systolic BP, diastolic BP and heart rate will be flagged with an "I" (increase) or "D" (decrease), respectively. If applicable, data from unscheduled vital signs assessments will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics.

In addition, a separate listing of all vital signs data outside their reference ranges by subject will also be provided.

The reference ranges (from the Quotient SOP "The Interpretation of the Electrocardiogram, Vital Signs and Clinical Laboratory Data During Phase I / II Clinical Trials") defined in Table 4 will be used.

Table 4 Vital Signs Reference Ranges

| Parameter | Split | Lower limit | Upper limit |
|-----------------------|-------------|-------------|-------------|
| Systolic BP | 18-45 years | 90 mmHg | 140 mmHg |
| Systolic BP | >45 years | 90 mmHg | 160 mmHg |
| Diastolic BP | NA | 40 mmHg | 90 mmHg |
| Heart rate | NA | 40 bpm | 100 bpm |
| Oral Body Temperature | NA | 35.5°C | 37.5°C |

NA=Not applicable

#### 10.6 ECGs

The details of measurement of supine ECG parameters (ie ventricular rate, QT interval, QTcF interval, PR interval, QRS duration, QRS axis and interpretation) are described in the study protocol. ECG parameters will be reported in the order given above in both summary tables and data listings.

#### 10.6.1 Summary Tables for ECGs

ECG data, including change from baseline (Day 1, Pre-dose for each study part), will be summarised (ie n, mean, SD, median, minimum and maximum) at each post-baseline time point by study part. The number and percentage of subjects with normal and prolonged QT intervals corrected for heart rate using Fridericia's correction (ie QTcF) and increases in QTcF intervals from baseline within the categories defined in Table 5 (based on the International Council on Harmonisation [ICH] E14 guideline [1]) will be summarised by time point within each study part. Percentages will be based on the number of subjects with measurements at the relevant time point.

For 'Overall' counts the worst (highest) value for each subject will be used for the counts. For the parameter 'Increase in QTcF interval from baseline', decreases in QTcF value fall into the <30 category (ie every subject should appear once in this summary table and actual change rather than absolute change is used for this parameter).

Table 5 ICH E14 Ranges for QTcF Intervals

| Parameter | ICH E14 Range |
|--------------------------------------------|---------------|
| | ≤450 msec |
| QTcF intervals | 451-480 msec |
| QTO Intervals | 481-500 msec |
| | >500 msec |
| | <30 msec |
| Increase in QTcF interval from<br>baseline | 30-60 msec |
| | >60 msec |

#### 10.6.2 Listings for ECGs

All ECG measurements (ie single readings), including derivations such as change from baseline, will be listed.

All ECG measurements will be flagged with an "H" or an "L" for values that are higher or lower than their reference ranges, respectively. If applicable, data from unscheduled ECG assessments will also be listed and flagged with a "#" to indicate it will not be used in the summary statistics.

In addition, subjects with increase in QTcF interval from baseline (30-60 msec) and with 'substantial increases' (>60 msec) will be flagged with 'l' and 'Sl', respectively.

A separate listing of all ECG parameters outside their reference range by subject will also be provided.

The reference ranges (from the Quotient SOP "The Interpretation of the Electrocardiogram, Vital Signs and Clinical Laboratory Data During Phase I / II Clinical Trials") and defined in Table 6 will be used.

Table 6 ECG Reference Ranges

| Parameter | Split | Lower limit | Upper limit |
|-----------------------|-------|-------------|-------------|
| Ventricular Rate (HR) | NA | 40 bpm | 100 bpm |
| QT Interval | NA | NA | 500 msec |
| QTcF Interval | Male | NA | 450 msec |
| PR Interval | NA | 120 msec | 220 msec |
| QRS Duration | NA | NA | 120 msec |
| QRS Axis | NA | -30° | 100° |

HR=heart rate
NA=Not applicable

#### 10.7 Body Weight

All body weight data will be listed. Body weight data from screening will be captured with demographic and baseline characteristics. Body weight data from admission to Part 2 will be listed separately.

#### 10.8 Physical Examination

All physical examination details and comments on any physical examination findings will be listed by subject for all subjects. Subjects who have no clinically significant findings at post treatment time points will be reported as 'No Clinically Significant Abnormal Findings' for the purposes of the listing.

# 11 Interim Statistical Analyses

No interim statistical analysis is planned for this study.

# 12 Changes in the Conduct of the Study or Planned Analysis

#### 12.1 Changes in the Conduct of the Study

No changes in the conduct of the study had been reported at the time this document was written.

#### 12.2 Changes to the Planned Analyses

For consistency across study parts, the definition of Tlag in part 2 was updated to match that of Tlag in Part 1. In addition, the definition of AUCextrap has been clarified.

#### 12.3 Any Other Relevant Changes

Not applicable.

#### 13 Overall Considerations

#### 13.1 Statistical Programming and Analysis

The Data Sciences Department at Quotient will perform the statistical programming and analysis to produce all analysis datasets and TFLs using the statistical SAS Software v9.4.

In general terms, categorical data will be presented using counts and percentages, whilst continuous variables will be presented using the n, mean, SD, median, minimum and maximum. For PK data, additional statistics including CV%, geometric n, geometric mean, geometric SD and geometric CV% will be presented, as appropriate. The geometric n is the

number of subjects included in the calculation of the geometric mean, geometric SD and geometric CV%.

The geometric mean is obtained by applying a natural log transformation to the raw data, calculating the arithmetic mean of the transformed values and then back transforming the arithmetic mean.

The following formula will be used to calculate the geometric SD:

ie a natural log transformation is applied to the raw data, the arithmetic SD of the transformed values is calculated, and then the arithmetic SD of the transformed values is back transformed.

The following formula will be used to calculate the geometric CV%:

geometric CV% = 
$$100 \times (exp{SD[log(raw data)]}^{2}-1)^{1/2}$$

ie a natural log transformation is applied to the raw data, the arithmetic SD of the transformed values is calculated. This value is then squared. The square value is back transformed and a value of 1 is subtracted from the back transformed value. A square root is then applied and the resulting value is multiplied by 100.

In general, summary statistics will be presented as detailed in Table 7 below, unless otherwise stated:

**Table 7 Reporting Conventions for Summary Statistics** 

| Data Type | Statistic | Number of decimal places for reporting (i) |
|---|---|---|
| Frequency Count | Counts (n) | None |
| | Percentages (%) | 1 decimal place |
| Summary statistic | n | None |
| | Mean | i + 1 decimal places |
| | Median | i + 1 decimal places |
| | SD | i + 1 decimal places |
| | Min | i decimal places |
| | Max | i decimal places |
| | CV% | 1 decimal place |
| | Geometric n | None |
| | Geometric Mean | i + 1 decimal places |
| | Geometric SD | i + 1 decimal places |
| | Geometric CV% | 1 decimal place |

i refers to the number of decimal places reported in the database or other appropriate source data for the original data

Note: The above table relates to rounding of summary stats from data received to certain number of decimal places. Summary stats on data received to a certain number of significant figures will be presented to the same number of significant figures as the data.

Details of how the PK parameters will be presented are detailed in Section 9.1.1. Where data requires rounding, values ending with 1 to 4 will be rounded down and values ending with 5 to 9 will be rounded up.

All data listings will be based on all enrolled subjects (as defined in Section 3.2.1). Details of age and sex will be included on all data listings.
If any nominal baseline measurements are found to be missing then consideration will be given to imputation using the preceding time point (eg Screening, Admission, if applicable). Unscheduled assessment may be used if appropriate. Details of any such imputations will be documented as part of the safety population.

There will be no other imputations for the safety data with regard to missing values or study discontinuation (ie subjects who do not complete the study). Imputation for PK parameter estimation using WinNonlin is described in Section 9.1.2 and for mass balance parameter estimation using SAS Software is described in Section 9.3.2. Imputations for reporting PK are described in Section 9.2.1.

If partial dates are available for smoking history, prior medications or medical/surgical history, there will be no date imputations. The data listings will only show the date information for the date part that is available (eg if only the year part of the date is available then YYYY will be presented in the listing). If the full date information is missing, then this will be presented as missing on the data listing.

#### 13.2 Quality Control of Summary Tables, Figures and Listings

Isolated data errors detected as a result of the QC checks that are deemed significant (ie errors that would impact the interpretation of the results in relation to the study objectives) will be corrected as per the data management plan. Systematic data errors will be investigated further. The data will be corrected if necessary, and the appropriate table, figure, and/or listing re-generated and then re-checked.

In addition to QC checks, a documented peer review will be performed of all SAS Software-generated report standard summary tables, figures and data listings, including a review of SAS Software code and program log files.

#### 13.2.1 Quality Control - Summary Tables

Manual QC methods (ie comparison of results in the table to results calculated by a calculator or spreadsheet) will be used for all summary tables. All summary tables will be QC'd as follows:

- for tables presented by study part only (ie no time points), all summary statistics will be OC'd
- for tables presented by study part and time point, at least one time point in each table will be QC'd – different combinations of time point will be selected across tables
- where tables are produced using a macro for multiple parameters, a minimum of 3 tables, using study part and time point as appropriate, will be QC'd
- for AEs, the study part/treatment details will be 100% QC'd against the treatment allocation list for all subjects
- AE summary tables will be 100% checked using the relevant data listing

#### 13.2.2 Quality Control - Figures

All figures will be QC'd manually using the corresponding/appropriate summary table or data listing, as follows:

- all data points for treatment will be checked
- where figures are produced using a macro for individual subjects and/or multiple parameters, a minimum of 3 figures will be QC'd
- mean figures will be QC'd using the corresponding summary table

### 13.2.3 Quality Control - Data Listings

All data listings will be subjected to a 100% manual QC check against the study database or other appropriate source data for a minimum of 2 subjects. If appropriate, the subjects checked will include at least one subject who withdrew early from the study.

#### 14 SAS Data Transfer

All SAS datasets used for analysis and reporting will be transferred to Kadmon on issue of the final CSR. This will be performed in compliance with CDISC ADaM (IG v1.1), data will be transferred as SAS Software transport files and will include define.xml (v2.0) output as well as a Data Reviewers Guide in pdf, which will be linked to the ADaM define.xml.

In addition, KD025m1 and KD025m2 Part 1 data provided by Covance will not be reported or analysed but will be transferred to Kadmon as raw data and will be included in the SDTM datasets

### 15 Programming Conventions

Quotient standards for layout of tables, figures and data listings and programming conventions will be used as follows:

- courier new, font size 8
- landscape
- US letter size (8.5 x 11 inches)

Tables and listings will be produced as MS Word 2016 documents and figures will be produced as PDF files. Listings will be sorted by subject ID number and treatment (where applicable).

The mock tables (Section 20) presented are a representation of Quotient reporting standards. However these are provided for illustrative purposes only. The numbering and titles of all TFLs and the formatting, labelling, footnotes and cosmetic appearance of tables may be modified or additional labelling/footnotes may need to be added during analysis and reporting, for clarification purposes. Any such changes will not be regarded as changes to planned analyses.

#### 16 Reference List

[1] International Council for Harmonisation (ICH) Topic E 14, The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs Guidelines approved by the Committee for Medicinal Products for Human Use (CHMP) in May 2005 which came into force November 2005.

## 17 Index of Tables

| Table<br>Number | Table Title |
|---|---|
| | Subject Disposition, Populations and Datasets |
| 14.1.1 | Subject Disposition by Reason<br>Summary Statistics: All Enrolled Subjects<br>Part 1 & Part 2 |
| 14.1.2.1 | Analysis Populations<br>Summary Statistics: All Enrolled Subjects<br>Part 1 & Part 2 |
| 14.1.2.2 | Analysis Datasets Summary Statistics: PK Population Part 1 & Part 2 |
| | (Programming note: Only produce table if there is a PK analysis dataset. If no PK or mass balance analysis dataset defined then do not produce table 14.1.2.2 or 14.1.2.3, and re-number table 14.1.2.1 as 14.1.2) |
| 14.1.2.3 | Analysis Datasets Summary Statistics: Mass Balance Population Part 1 & Part 2 |
| | (Programming note: Only produce table if there is a mass balance analysis dataset defined. If no PK or mass balance dataset defined then do not produce table 14.1.2.2 or 14.1.2.3, and re-number table 14.1.2.1 as 14.1.2. If there is a mass balance dataset but no PK dataset, then do not produce table 14.1.2.2 and re-number table 14.1.2.3 as 14.1.2.2) |
| | Demographic and Baseline Characteristics |
| 14.1.3 | Demographic and Baseline Characteristics Summary Statistics: Safety Population Part 1 & Part 2 |
| 14.1.4 | Lifestyle Details: Smoking History and Alcohol Consumption at Baseline Summary Statistics: Safety Population Part 1 & Part 2 |
| | Dosing Details |
| 14.1.5.1 | Extent of Exposure Summary Statistics: Safety Population Part 1 |
| 14.1.5.2 | Extent of Exposure Summary Statistics: Safety Population Part 2 |
| | Plasma and Whole Blood Pharmacokinetic Concentrations |

| Table<br>Number | Table Title |
|---|---|
| 14.2.1.1 | Plasma Pharmacokinetic Concentrations Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 1: KD025 Oral Tablet &amp; [14C]-KD025 IV Infusion <kd025 (units)="" [14c]-kd025=""></kd025></pk> |
| 14.2.1.2.1 | Plasma Pharmacokinetic Concentrations Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <kd025 (units)="" kd025m1="" kd025m2=""></kd025></pk> |
| 14.2.1.2.2 | Plasma Pharmacokinetic Concentrations: Total Radioactivity Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule</pk> |
| 14.2.1.2.3 | Whole Blood Pharmacokinetic Concentrations: Total Radioactivity Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule</pk> |
| 14.2.1.2.4 | Whole Blood:Plasma Concentration Ratios: Total Radioactivity Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule</pk> |
| | Plasma and Whole Blood Pharmacokinetic Parameters |
| 14.2.2.1 | Plasma Pharmacokinetic Parameters Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 1: KD025 Oral Tablet &amp; [14C]-KD025 IV Infusion &lt; KD025 / [14C]-KD025 &gt;</pk> |
| 14.2.2.2.1 | Plasma Pharmacokinetic Parameters Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule &lt; KD025 / KD025m1 / KD025m2 &gt;</pk> |
| 14.2.2.2.2 | Plasma Pharmacokinetic Parameters: Total Radioactivity Summary Statistics: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule</pk> |
| 14.2.2.2.3 | Whole Blood Pharmacokinetic Parameters: Total Radioactivity Summary Statistics: < <i>PK Population/PK Analysis Dataset&gt;</i> Part 2: [14C]-KD025 Oral Capsule |
| 14.2.2.3 | Relative Bioavailability of Oral Formulations: KD025<br>Summary Statistics: <pk analysis="" dataset="" pk="" population=""><br/>Part 1 &amp; Part 2</pk> |
| ; | Excretion and Recovery – Urine Concentrations |
| 14.2.3.1.1 | Excretion: Total Radioactivity Ae(Urine) by Collection Period < Units> Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |

| Table<br>Number | Table Title |
|---|---|
| 14.2.3.1.2 | Excretion: Total Radioactivity Cumulative Ae(Urine) < Units > Summary Statistics: < Mass Balance Population/Mass Balance Analysis Dataset > Part 2: [14C]-KD025 Oral Capsule |
| 14.2.3.1.3 | Recovery: Total Radioactivity %Ae(Urine) by Collection Period Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| 14.2.3.1.4 | Recovery: Total Radioactivity Cumulative %Ae(Urine) Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| | Excretion and Recovery – Faécal Concentrations |
| 14.2.3.2.1 | Excretion: Total Radioactivity Ae(Faeces) by Collection Period < <i>Units&gt;</i> Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| 14.2.3.2.2 | Excretion: Total Radioactivity Cumulative Ae(Faeces) < Units> Summary Statistics: < Mass Balance Population/Mass Balance Analysis Dataset> Part 2: [14C]-KD025 Oral Capsule |
| 14.2.3.2.3 | Recovery: Total Radioactivity %Ae(Faeces) by Collection Period Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| 14.2.3.2.4 | Recovery: Total Radioactivity Cumulative %Ae(Faeces) Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| | Excretion and Recovery – Urine and Faeces Combined |
| 14.2.3.3.1 | Excretion: Total Radioactivity Ae(Total) by Collection Period < <i>Units</i> > Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |

| Table<br>Number | Table Title |
|---|---|
| 14.2.3.3.2 | Excretion: Total Radioactivity Cumulative Ae(Total) < Units> Summary Statistics: < Mass Balance Population/Mass Balance Analysis Dataset> Part 2: [14C]-KD025 Oral Capsule |
| 14.2.3.3.3 | Recovery: Total Radioactivity %Ae(Total) by Collection Period Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| 14.2.3.3.4 | Recovery: Total Radioactivity Cumulative %Ae(Total) Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| | Cumulative Excretion and Recovery Parameters |
| 14.2.3.4 | Excretion and Recovery: Total Radioactivity Overall Cumulative Excretion and Recovery Parameters Summary Statistics: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| | Adverse Events |
| 14.3.1.1 | Overall Summary of Treatment-Emergent Adverse Events Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.3.1.2 | Subjects Reporting Treatment-Emergent Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.3.1.3 | Subjects Reporting Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Severity Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.3.1.4 | Subjects Reporting Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Relationship to IMP Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.3.1.5 | Subjects Reporting Adverse Drug Reactions By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |

| Table<br>Number | Table Title |
|---|---|
| 14.3.1.6 | Subjects Reporting Serious Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.3.2.1 | Overall Summary of Treatment-Emergent Adverse Events Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.3.2.2 | Subjects Reporting Treatment-Emergent Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.3.2.3 | Subjects Reporting Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Severity Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.3.2.4 | Subjects Reporting Treatment-Emergent Adverse Events By MedDRA System Organ Class, Preferred Term and Relationship to IMP Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.3.2.5 | Subjects Reporting Adverse Drug Reactions By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.3.2.6 | Subjects Reporting Serious Adverse Events By MedDRA System Organ Class and Preferred Term Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| | Laboratory Results |
| 14.4.1.1 | Haematology Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.4.1.2 | Haematology Shift Table: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.4.1.3 | Clinical Chemistry Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.4.1.4 | Clinical Chemistry Shift Table: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |

| Table<br>Number | Table Title |
|---|---|
| 14.4.2.1 | Haematology Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.4.2.2 | Haematology Shift Table: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.4.2.3 | Clinical Chemistry Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.4.2.4 | Clinical Chemistry Shift Table: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| _ | Vital Signs and ECG Results |
| 14.5.1.1 | Vital Signs Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.5.1.2.1 | ECGs Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.5.1.2.2 | ECGs QTcF Categorical Data Summary Statistics: Safety Population Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 14.5.2.1 | Vital Signs Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.5.2.2.1 | ECGs Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |
| 14.5.2.2.2 | ECGs QTcF Categorical Data Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule |

18 Index of Figures

| Figure<br>Number | Figure Title |
|---|---|
| | Whole Blood and Plasma Pharmacokinetic Concentrations |
| 14.2.2.1.1 | Plasma Pharmacokinetic Concentrations Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: < <i>PK Population/PK Analysis Dataset&gt;</i> Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion < <i>KD025 / [14C]-KD025 &gt;</i> |
| 14.2.2.1.2 | Plasma Pharmacokinetic Concentrations Log10/Linear Scale Geometric Mean (×/÷ Geometric SD) Values: < <i>PK Population/PK Analysis Dataset&gt;</i> Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion < KD025 / [14C]-KD025 > |
| 14.2.2.1.3 | Plasma Pharmacokinetic Concentrations Linear/Linear Scale Spaghetti Plots of All Individual Values: < PK Population/PK Analysis Dataset> Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion < KD025 / [14C]-KD025 > |
| 14.2.2.1.4 | Plasma Pharmacokinetic Concentrations Log10/Linear Scale Spaghetti Plots of All Individual Values: < PK Population/PK Analysis Dataset> Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion < KD025 / [14C]-KD025 > |
| 14.2.2.2.1 | Plasma Pharmacokinetic Concentrations Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: < <i>PK Population/PK Analysis Dataset&gt;</i> Part 2: [14C]-KD025 Oral Capsule (Programming note: KD025, KD025m1, KD025m2 and total radioactivity will be overlaid on the same plot) |
| 14.2.2.2,2 | Plasma Pharmacokinetic Concentrations Log10/Linear Scale Geometric Mean (×/÷ Geometric SD) Values: < <i>PK Population/PK Analysis Dataset&gt;</i> Part 2: [14C]-KD025 Oral Capsule |
| | (Programming note: KD025. KD025m1, KD025m2 and total radioactivity will be overlaid on the same plot) |

| Figure<br>Number | Figure Title |
|---|---|
| 14.2.2.2.3 | Plasma and Whole Blood Pharmacokinetic Concentrations: Total Radioactivity Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: < <i>PK Population/PK Analysis Dataset</i> > Part 2: [14C]-KD025 Oral Capsule (Programming note: Plasma and whole blood total radioactivity |
| 14.2.2.2.4 | concentrations will be overlaid on the same plot) Plasma and Whole Blood Pharmacokinetic Concentrations: Total Radioactivity Log10/Linear Scale Geometric Mean (×/÷ Geometric SD) Values: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule (Programming note: Plasma and whole blood total radioactivity</pk> |
| 14.2.2.2.5 | concentrations will be overlaid on the same plot) Plasma Pharmacokinetic Concentrations Linear/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <analyte> (Programming note: KD025, KD025m1 and KD025m2 will be displayed on separate pages)</analyte></pk> |
| 14.2.2.2.6 | Plasma Pharmacokinetic Concentrations Log10/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <analyte> (Programming note:KD025, KD025m1 and KD025m2 will be displayed on separate pages)</analyte></pk> |

| Figure<br>Number | Figure Title |
|---|---|
| 14.2.2.2.7 | Plasma and Whole Blood Pharmacokinetic Concentrations: Total Radioactivity Linear/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <plasma blood="" radioactivity="" total="" whole=""> (Programming note: Plasma and whole blood total radioactivity will be displayed on separate pages)</plasma></pk> |
| 14.2.2.2.8 | Plasma and Whole Blood Pharmacokinetic Concentrations: Total Radioactivity Log10/Linear Scale Spaghetti Plots of All Individual Values: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <plasma blood="" radioactivity="" total="" whole=""> (Programming note: Plasma and whole blood total radioactivity will be displayed on separate pages)</plasma></pk> |
| 14.2.2.2.9 | Plasma and Whole Blood Pharmacokinetic Concentrations Linear/Linear Scale Individual Values for Subject <xxx>: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <subject> (Programming note: KD025, KD025m1, KD025m2 and total radioactivity [plasma and whole blood] will be overlaid on the same plot)</subject></pk></xxx> |
| 14.2.2.2.10 | Plasma and Whole Blood Pharmacokinetic Concentrations Log10/Linear Scale Individual Values for Subject <xxx>: <pk analysis="" dataset="" pk="" population=""> Part 2: [14C]-KD025 Oral Capsule <subject> (Programming note: KD025, KD025m1, KD025m2 and total radioactivity [plasma and whole blood] will be overlaid on the same plot)</subject></pk></xxx> |

| Figure<br>Number | Figure Title |
|---|---|
| 14.2.2.3.1 | Plasma Pharmacokinetic Concentrations: Oral Formulations, KD025 Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: <pk analysis="" dataset="" pk="" population=""> Part 1 and 2 (Programming note: Treatments A and C will be overlaid on the same plot)</pk> |
| 14.2.2.3.2 | Plasma Pharmacokinetic Concentrations: Oral Formulations, KD025 Log10/Linear Scale Geometric Mean (×/÷Geometric SD) Values: < <i>PK Population/PK</i> Analysis Dataset> Parts 1 and 2 (Programming note: Treatments A and C will be overlaid on the same plot) |
| , | Cumulative Excretion and Recovery |
| 14.2.3.1 | Mean Cumulative Excretion of Total Radioactivity CumAe(Urine), CumAe(Faeces) and CumAe(Total) Linear/Linear Scale Arithmetic Mean (± Arithmetic SD) Values: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |
| 14.2.3.2 | Mean Cumulative Recovery of Total Radioactivity Cum%Ae(Urine), Cum%Ae(Faeces) and Cum%Ae(Total) Linear/Linear Scale Arithmetic Mean (±Arithmetic SD) Values: <mass analysis="" balance="" dataset="" mass="" population=""> Part 2: [14C]-KD025 Oral Capsule</mass> |

# 19 Index of Listings

| Listing<br>Number | Listing Title |
|---|---|
| | Subject Informed Consent and Completion/Withdrawal |
| 16.2.1 | Subject Informed Consent and Completion/Withdrawal Individual Values: All Enrolled Subjects Part 1 & Part 2 |
| , | Protocol Deviations and Inclusion/Exclusion Criteria |
| 16.2.2.1 | Protocol Deviations<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.2.2 | Inclusion/Exclusion Criteria Individual Values: All Enrolled Subjects Part 1 & Part 2 |
| | Analysis Populations and Reasons for Exclusion |
| 16.2.3.1 | Analysis Populations and Reasons for Exclusion Individual Values: All Enrolled Subjects Part 1 & Part 2 |
| | (Programming note: If analysis datasets are not required, then this listing will be re-numbered from 16.2.3.1 to 16.2.3 and Listing 16.2.3.2 will not be produced) |
| 16.2.3.2 | Analysis Datasets and Reasons for Exclusion Individual Values: All Enrolled Subjects Part 1 & Part 2 |
| | (Programming note: If analysis datasets are not required, then this listing will not be produced and Listing 16.2.3.1 will be re-numbered from 16.2.3.1 to 16.2.3) |
| | Demographic and Baseline Characteristics |
| 16.2.4.1 | Demographics and Baseline Characteristics<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.4.2 | Lifestyle Details: Smoking History and Alcohol Consumption Individual Values: All Enrolled Subjects Part 1 & Part 2 |
| 16.2.4.3 | Medical/Surgical History<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.4.4 | Prior and Concomitant Medication<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.4.5 | Urine Drug Screen<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.4.6 | Alcohol Breath and Carbon Monoxide Breath Test<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.4.7 | Virology<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.4.8 | Creatinine Clearance<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| , | Dosing Details and Meal Details |
| 16.2.5.1.1 | Dosing Details<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| 16.2.5.1.2 | Meal Details<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |
| | Urine and Faecal Concentration Data |
| 16.2.5.2.1 | Urine Collection and Weight Details<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.5.2.2 | Urine Concentrations, Excretion and Recovery: Total Radioactivity (units) Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.5.2.3 | Faecal Collection and Weight Details<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.5.2.4 | Faecal Concentrations, Excretion and Recovery: Total Radioactivity (units) Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.5.2.5 | Total Urine and Faecal Concentrations, Excretion and Recovery: Total Radioactivity (units) Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| | Plasma and Whole Blood Pharmacokinetic Concentration Data |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.5.3.1.1 | Blood Sample Collection Details for Pharmacokinetic Analysis Individual Values: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.5.3.1.2 | Plasma Pharmacokinetic Concentrations Individual Values: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion < KD025 / [14C]-KD025 > |
| 16.2.5.3.2.1 | Blood Sample Collection Details for Pharmacokinetic Analysis Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.5.3.2.2 | Plasma Pharmacokinetic Concentrations Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule < KD025 / KD025m1 / KD025m2 > |
| 16.2.5.3.2.3 | Plasma and Whole Blood Pharmacokinetic Concentrations: Total Radioactivity Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule (Programming note: This listing will include whole blood:plasma concentration ratios) |
| | Plasma and Whole Blood Pharmacokinetic Parameter Data |
| 16.2.6.1.1 | Plasma Pharmacokinetic Parameters Individual Values: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion < KD025 / [14C]-KD025 > |
| 16.2.6.2.1 | Plasma Pharmacokinetic Parameters Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule < KD025 / KD025m1 / KD025m2 > |
| 16.2.6.2.2 | Plasma and Whole Blood Pharmacokinetic Parameters: Total Radioactivity Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule <plasma blood="" whole=""></plasma> |
| 16.2.6.3 | Relative Bioavailability of Oral Formulations, KD025<br>Individual Values: All Enrolled Subjects<br>Part 1 & Part 2 |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.6.4 | Pharmacokinetic Parameter Flags |
| | (Programming note: Details of the PK parameter flags will be added to listing 16.2.6.1.1 and 16.2.6.2.1 as footnotes if length of these details allows – in which case do not produce this listing. Otherwise display PK parameter flags in this listing) |
| | Adverse Events |
| 16.2.7.1.1 | Pre-dose Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.7.1.2 | All Treatment-Emergent Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.7.1.3 | Serious Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.7.2.1 | Pre-dose Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.7.2.2 | All Treatment-Emergent Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.7.2.3 | Serious Adverse Events<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| | Laboratory Data |
| 16.2.8.1.1.1 | Blood Sample Collection Details for Laboratory Analysis Individual Values: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.1.2 | Blood Sample Collection Comments Individual Values: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.2.1 | Haematology<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.2.2 | Haematology<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.3.1 | Clinical Chemistry<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |

| Listing<br>Number | Listing Title |
|---|---|
| 16.2.8.1.3.2 | Clinical Chemistry Individual Values Outside the Reference Range: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.4.1 | Urinalysis Sample Collection<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.4.2 | Urinalysis<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.1.4.3 | Urinalysis Individual Values Outside the Reference Range: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.8.2.1.1 | Blood Sample Collection Details for Laboratory Analysis<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.1.2 | Blood Sample Collection Comments Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.2.1 | Haematology<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.2.2 | Haematology<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.3.1 | Clinical Chemistry Individual Values: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.3.2 | Clinical Chemistry Individual Values Outside the Reference Range: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.4.1 | Urinalysis Sample Collection<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.4.2 | Urinalysis<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.8.2.4.3 | Urinalysis Individual Values Outside the Reference Range: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |

| Listing<br>Number | Listing Title |
|---|---|
| | Vital Signs and ECGs |
| 16.2.9.1.1.1 | Vital Signs<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.9.1.1.2 | Vital Signs Individual Values Outside the Reference Range: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.9.1.2.1 | ECGs<br>Individual Values: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| | (Programming note: The order of ECG parameters is to be as per Section 10.6) |
| 16.2.9.1.2.2 | ECGs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.9.2.1.1 | Vital Signs<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.9.2.1.2 | Vital Signs Individual Values Outside the Reference Range: All Enrolled Subjects Part 2: [14C]-KD025 Oral Capsule |
| 16.2.9.2.2.1 | ECGs<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| | (Programming note: The order of ECG parameters is to be as per Section 10.6) |
| 16.2.9.2.2.2 | ECGs<br>Individual Values Outside the Reference Range: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| | Other Data |
| 16.2.9.3.1 | Physical Examination Data Individual Values: All Enrolled Subjects Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion |
| 16.2.9.3.2.1 | Physical Examination Data<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |
| 16.2.9.3.2.2 | Body Weight Data<br>Individual Values: All Enrolled Subjects<br>Part 2: [14C]-KD025 Oral Capsule |

| Sponsor | r/Quotient | Sciences | Confidentia | ı |
|---------|------------|----------|-------------|---|

20 Mock Tables

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.1

Subject Disposition by Reason

Summary Statistics: All Enrolled Subjects

Part 1 & Part 2

| | OVERALL (N=X) n (%) |
|-------------------------------------------|---------------------|
| Subjects enrolled (1) | xx (xx.x) |
| Subjects dosed | |
| in Part 1 | xx (xx.x) |
| in Part 2 | xx (xx.x) |
| Subjects completed | xx (xx.x) |
| Subjects discontinued | xx (xx.x) |
| Reason for discontinuation | |
| REASON 1 | xx (xx.x) |
| REASON 2 | xx (xx.x) |
| REASON 3 | xx (xx.x) |
| *** | *** |
| <all categories="" on="" source=""></all> | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 and a 200 mg KD025 oral capsule in Part 2

A subject may be discontinued for one reason only. (1) An enrolled subject signed the informed consent, qualified per the inclusion/exclusion criteria and was allocated a subject number

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all reasons for discontinuation as recorded

on the source. If none of the subjects discontinued from the study early

then reasons for discontinuation will not be populated in the summary table

Programming note: Percentages are based on the number of subjects enrolled

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.2.1
Analysis Populations

Summary Statistics: All Enrolled Subjects

Part 1 & Part 2

| | Part 1<br>(N=X)<br>n (%) | Part 2<br>(N=X)<br>n (%) | OVERALL (N=X) n (%) |
|---|---|---|---|
| Number (%) of subjects in safety population<br>Reasons for exclusion from safety population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <all categories="" from="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number (%) of subjects in PK population Reasons for exclusion from PK population | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <all categories="" from="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number (%) of subjects in mass balance population Reasons for exclusion from mass balance population | | xx (xx.x) | xx (xx.x) |
| <all categories="" from="" source=""></all> | | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 and a 200 mg KD025 oral capsule in Part 2

A subject may be excluded for more than one reason

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all reasons for exclusion as recorded

on the source. If none of the subjects were excluded from a population

then reasons for exclusion will not be populated in the summary table.

Programming note: Percentages are based on the number of subjects enrolled

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.2.2
Analysis Datasets

Summary Statistics: PK Population

Part 1 & Part 2

| | Part 1<br>(N=X)<br>n (%) | Part 2<br>(N=X)<br>n (%) | OVERALL (N=X) n (%) |
|---|---|---|---|
| Number (%) of subjects in PK analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons for exclusion from PK analysis set<br><all categories="" from="" source=""></all> | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1

and a 200 mg KD025 oral capsule in Part 2

A subject may be excluded for more than one reason

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB\_XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all reasons for exclusion as recorded

on the source. If none of the subjects were excluded from an analysis set

then reasons for exclusion will not be populated in the summary table. Programming note: Repeat for mass balance population on separate page (with sub-heading

'Summary Statistics: Mass Balance Population') if required

Programming note: Produce similar table for mass balance population (if mass balance dataset defined)

as table 14.1.2.3 if a PK dataset is also defined or 14.1.2.2 if not.

Programming note: Percentages are based on the number of subjects in the relevant population

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.3

Demographic and Baseline Characteristics Summary Statistics: Safety Population

Part 1 & Part 2

| | | OVERALL<br>(N=X) |
|---|---|---|
| Age (years) | n<br>Mean<br>SD<br>Median<br>Min<br>Max | xx<br>xx.x<br>xx.x<br>xx.x<br>xx |
| Ethnicity n(%) | <all categories="" on="" source=""></all> | xx (xx.x) |
| Race n(%) | <all categories="" on="" source=""></all> | xx (xx.x) |
| Sex n(%) | Male | xx (xx.x) |
| Height (cm) | <del></del> | |
| Weight (kg) | | ••• |
| BMI (kg/m^2) | | |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1 and a 200 mg KD025 oral capsule in Part 2

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will continue for all categories of ethnicity and race.

Height, Weight and BMI will be assessed using the same descriptive statistics as Age.

If any values are missing, then a "missing" row will be included in the table, as applicable

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.4

Lifestyle Details: Smoking History and Alcohol Consumption at Baseline

Summary Statistics: Safety Population

Part 1 & Part 2

| | | (N=X)<br>n (%) |
|---|---|---|
| Does subject smoke (1) | NO<br>PREVIOUSLY | xx (xx.x)<br>xx (xx.x) |
| Alcohol Consumption (2) | NONE YES: NOT REGULAR (2) | xx (xx.x)<br>xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 and a 200 mg KD025 oral capsule in Part 2

Baseline is defined as at Screening

(1) Anyone who smoked or used e-cigarettes or nicotine replacement products in the last 12 months is excluded from the study. (2) Anyone who regularly consumes alcohol (>21 units/week in males) is excluded from the study. 1 unit = 1/2 pint beer, 25 mL of 40% spirit, 1.5 to 2 units = 125 mL glass of wine depending on type

OVERALL

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB\_XX

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.5.1 Extent of Exposure

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

| 100 u | r [14C | 1-KD025 | IV | Infusion | (N=X) |
|-------|--------|---------|----|----------|-------|
|-------|--------|---------|----|----------|-------|

| | 200 mg KD025 Oral | 100 μg [110] ΚΕΟΣΟ | IV IIII usion (N-A) |
|-----------|-------------------|--------------------|---------------------|
| Statistic | Tablet (N=X) | (µg) | (kBq) |
| n | xx | xx | xx |
| Mean | | xx.xx | xx.xx |
| SD | | xx.xx | xx.xx |
| Median | | xx.xx | xx.xx |
| Min | | xx.x | xx.x |
| Max | | xx.x | xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB\_XX

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.1.5.2 Extent of Exposure

Summary Statistics: Safety Population Part 2: [14C]-KD025 Oral Capsule

200 mg [14C]-KD025 Oral Capsule (N=X)

| Statistic | (mg) | (MBq) | (µCi) |
|-----------|-------|-------|-------|
| n | xx | xx | xx |
| Mean | xx.xx | xx.xx | xx.xx |
| SD | xx.xx | xx.xx | xx.xx |
| Median | xx.xx | xx.xx | xx.xx |
| Min | xx.x | xx.x | xx.x |
| Max | xx.x | xx.x | xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg [14C]-KD025 oral capsule in Part 2

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.2.1.1

Plasma Pharmacokinetic Concentrations

Summary Statistics: <PK Population/PK Analysis Dataset>
Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

KD025 <units> (N=X)

| | | Arithmetic (1) | | | | | Geometric (2) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | 'n | Mean | SD | CV% | Median | Min | Max | n | Mean | SD | CV% |
| PRE-DOSE | xx | xx.xxx | xx.xxx | xx.x | xx.xxx | xx.xx | xx.xx | | | | |
| TIME POINT 1 | xx | xx.xxx | xx.xxx | xx.x | xx.xxx | xx.xx | xx.xx | xx | xx.xxx | xx.xxx | xx.x |
| TIME POINT 2 | xx | xx.xxx | xx.xxx | xx.x | xx.xxx | xx.xx | xx.xx | xx | xx.xx | xx.xxx | xx.x |
| TIME POINT 3 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.xx | xx.xx | xx | xx.xx | xx.xx | xx.x |
| *** | | ••• | ••• | ••• | | ••• | | ••• | ••• | ••• | ••• |
| <all other="" points="" time=""></all> | xx | xx.xxx | xx.xxx | xx.x | XX.XXX | xx.xx | XX.XX | xx | XX.XXX | XX.XXX | XX X |

Note: The data in this table are presented in listing x.x

- All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1 No imputation was carried out for concentration values reported as NR (not reportable/no result) or NS (no sample)
- The LLOQ value was <value, units>
  (1) For arithmetic summary statistics, concentration values reported as BLQ are set to zero.
- (2) Geometric summary statistics are not calculated for the pre-dose time-point. For calculation of geometric summary statistics, values reported as BLQ are set to ½ × LLOQ.

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all time points for each analyte on a new page Programming note: Similar tables will be produced for Part 2 (update heading and footnote accordingly) for:

- Table 14.2.1.2.1 ie Plasma Pharmacokinetic Concentrations
- Table 14.2.1.2.2 ie Plasma Pharmacokinetic Concentrations: Total Radioactivity
- Table 14.2.1.2.3 ie Whole Blood Pharmacokinetic Concentrations: Total Radioactivity

Page x of y

Kadmon Corporation LLC Protocol: KD025-108

TABLE 14.2.2.1

Plasma Pharmacokinetic Parameters

Summary Statistics: <PK Population/PK Analysis Dataset>
Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

KD025 (N=X)

PK Parameter

| Statistic | Parameter 1 (units) | Parameter 2 (units) | Parameter 3 (units) | | All Other PK Parameters<br>(units) |
|---|---|---|---|---|---|
| n | xx | xx | xx | ••• | xx |
| Mean | xx.xx | xx.xxx | xx.xxx | *** | xx.xx |
| SD | xx.xx | xx.xxx | xx.xxx | *** | xx.xxx |
| CV% | xx.x | xx.x | xx.x | *** | xx.x |
| Median | xx.xx | xx.xxx | xx.xxx | ••• | xx.xxx |
| Min | xx.xx | xx.xx | xx.xx | *** | xx.xx |
| Max | xx.xx | xx.xx | xx.xx | *** | xx.xx |
| Geometric n | xx | xx | xx | *** | xx |
| Geometric Mean | xx.xx | xx.xxx | xx.xxx | *** | xx.xxx |
| Geometric SD | xx.xx | xx.xxx | xx.xx | *** | xx.xx |
| Geometric CV% | xx.x | xx.x | xx.x | ••• | xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 The LLOQ value was <value, units>

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all parameters for each analyte on a new page Programming note: Similar tables will be produced for Part 2 (update heading and footnote accordingly) for:

- Table 14.2.2.2.1 ie Plasma Pharmacokinetic Parameters
- Table 14.2.2.2.2 ie Plasma Pharmacokinetic Parameters: Total Radioactivity
- Table 14.2.2.3 ie Whole Blood Pharmacokinetic Parameters: Total Radioactivity
- · Table 14.2.2.2.4 ie Whole Blood: Plasma Concentration Ratios: Total Radioactivity

Programming note: Similar tables will be produced without part and analyte headings (update footnote accordingly) for:

• Table 14.2.2.3 ie Relative Bioavailability of Oral Formulations: KD025

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.2.3.1.1

Excretion: Total Radioactivity

Ae(Urine) by Collection Period <(units)>

Summary Statistics: <Mass Balance Population/Mass Balance Analysis Dataset>

Part 2: [14C]-KD025 Oral Capsule

[14C]-KD025 (N=X)

| Collection Period | n | Mean | SD | CV% | Median | Min | Max |
|---|---|---|---|---|---|---|---|
| TIMEO-TIME1 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x |
| TIME1-TIME2 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x |
| TIME2-TIME3 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x |
| <all intervals="" other="" time=""></all> | <br>XX | **** | **** | | | | |
| ANTE OFFICE CIME INCOLVATOR | ^^ | XX.XX | xx.xx | XX.X | xx.xx | XX.X | XX.X |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg [14C]-KD025 oral capsule in Part 2

Where a subject has failed to void or has a BLQ concentration over a particular collection interval, the amount excreted (Ae) has been set to zero

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming Note: similar tables will be produced for:

- Table 14.2.3.1.3 ie %Ae(Urine) (Recovery)
- Table 14.2.3.2.1 ie Ae(Faeces)
- Table 14.2.3.2.3 ie %Ae(Faeces) (Recovery)
- Table 14.2.3.3.1 ie Ae[total]
- Table 14.2.3.3.3 ie %Ae[total] (Recovery)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.2.3.1.2

Excretion: Total Radioactivity Cumulative Ae(Urine) <(units)>

Summary Statistics: <Mass Balance Population/Mass Balance Analysis Dataset>

Part 2: [14C]-KD025 Oral Capsule

[14C]-KD025 (N=X)

| Collection Period | n | Mean | SD | CA% | Median | Min | Max |
|---|---|---|---|---|---|---|---|
| TIMEO-TIME1 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x |
| TIMEO-TIME2 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x |
| TIMEO-TIME3 | xx | xx.xx | xx.xx | xx.x | xx.xx | xx.x | xx.x |
| <all intervals="" other="" time=""></all> | <br>xx | <br>xx.xx | <br>xx.xx | <br>xx.x | <br>xx.xx | <br>XX.X | <br>xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg [14C]-KD025 oral capsule in Part 2

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: If required as a result of early withdrawal or varying follow-up periods, a further set of tables will be produced for LOCF values. Table numbers will be incremented by .1 for observed values and .2 for LOCF.

Programming note: Similar tables will be produced for:

- Table 14.2.3.1.4 ie Cumulative %Ae(Urine) (Recovery)
- Table 14.2.3.2.2 ie Cumulative Ae(Faeces)
- Table 14.2.3.2.4 ie Cumulative %Ae(Faeces) (Recovery)
- Table 14.2.3.3.2 ie Cumulative Ae[total]
- Table 14.2.3.3.4 ie Cumulative %Ae[total] (Recovery)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.2.3.4

Excretion and Recovery: Total Radioactivity

Overall Cumulative Excretion and Recovery Parameters

Summary Statistics: <Mass Balance Population/Mass Balance Analysis Dataset>

Part 2: [14C]-KD025 Oral Capsule

[14C]-KD025 (N=X)

| | Ur | Urine | | ces | Total | |
|---|---|---|---|---|---|---|
| | CumAe<br>(units) | Cum%Ae<br>(%) | CumAe<br>(units) | Cum%Ae<br>(%) | CumAe<br>(units) | Cum%Ae<br>(%) |
| n | xx | xx | xx | xx | xx | xx |
| Mean | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| CV% | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Median | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Min | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Max | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg [14C]-KD025 oral capsule in Part 2

CumAe represent cumulative excretion. Cum%Ae represents cumulative recovery as a percentage of the radioactive dose administered

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB\_XX

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.3.1.1

Overall Summary of Treatment-Emergent Adverse Events

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100 µg [14C]-KD025 IV infusion (N=X)

| Event | n(%) | Total Number<br>of Events |
|------------------------------------|-----------|---------------------------|
| TEAE | xx (xx.x) | xx |
| ADR (1) | xx (xx.x) | xx |
| Severe TËAE | xx (xx.x) | xx |
| Serious TEAE | xx (xx.x) | xx |
| TEAE leading to subject withdrawal | xx (xx.x) | xx |
| TEAE leading to death | xx (xx.x) | xx |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 TEAEs are coded using MedDRA v22.0

- (1) An ADR is any AE that the investigator considers possibly related or related to the IMP n is the number of subjects reporting at least one event
- PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: Similar table will be produced for Part 2 (ie Table 14.3.2.1)

Page x of y

TABLE 14.3.1.2

Subjects Reporting Treatment-Emergent Adverse Events

By MedDRA System Organ Class and Preferred Term

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu$ g [14C]-KD025 IV infusion (N=X)

| | • | |
|--------------------------|-----------|-------------|
| | n(%) | Events<br>n |
| Subjects Reporting TEAEs | xx (xx.x) | xx |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx |
| PREFFERED TERM 1 | xx (xx.x) | xx |
| PREFFERED TERM 2 | xx (xx.x) | xx |
| etc | ••• | |
| YSTEM ORGAN CLASS 2 | xx (xx.x) | xx |
| PREFFERED TERM 1 | xx (xx.x) | xx |
| PREFFERED TERM 2 | xx (xx.x) | xx |
| etc | *** | |
| • | ••• | *** |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1 TEAEs are coded using MedDRA v22.0 and are presented in descending order of frequency Subjects experiencing more than 1 episode of a TEAE are counted only once within each SOC and PT Event is the total number of TEAEs within the relevant SOC and PT

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: Counts of number of subjects are by maximum severity (ie using the most severe episode)

Programming note: Similar table will be produced for Part 2 (ie Table 14.3.2.2)

Page x of y

TABLE 14.3.1.3
Subjects Reporting Treatment-Emergent Adverse Events
By MedDRA System Organ Class, Preferred Term and Severity
Summary Statistics: Safety Population
Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100 µg [14C]-KD025 IV infusion (N=X)

| | | iild<br>(%) | | lerate<br>1(%) | | evere |
|---|---|---|---|---|---|---|
| Subjects Reporting TEAEs | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| SYSTEM ORGAN CLASS 1 | xx | (xx.x) | · xx | (xx.x) | xx | (xx.x) |
| PREFFERED TERM 1 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| PREFFERED TERM 2 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| etc | | | | ••• | | |
| SYSTEM ORGAN CLASS 2 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| PREFFERED TERM 1 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| PREFFERED TERM 2 | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) |
| etc | | ••• | | ••• | | |
| <b></b> | | ••• | | | | ••• |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1

TEAEs are coded using MedDRA v22.0 and are presented in descending order of frequency

Counts are given for total number of subjects, not for events

Counts of number of subjects are by maximum severity (ie subjects experiencing more than 1 episode

of a TEAE are counted only once within each SOC and PT using the most severe episode)

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX DDMMMYYYY HH:MM

Programming note: Similar table will be produced for Part 2 (ie Table 14.3.2.3)

Page x of y

TABLE 14.3.1.4

Subjects Reporting Treatment-Emergent Adverse Events

By MedDRA System Organ Class, Preferred Term and Relationship to IMP

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu$ g [14C]-KD025 IV infusion (N=X)

| | Unrelated Possibly Related n(%) n(%) | | Related<br>n(%) |
|---|---|---|---|
| Subjects Reporting TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PREFFERED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PREFFERED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc | *** | ••• | *** |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PREFFERED TERM 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PREFFERED TERM 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc | ••• | *** | ••• |
| | ••• | | *** |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100 µg [14C]-KD025 IV infusion in Part 1

TEAEs are coded using MedDRA v22.0 and are presented in descending order of frequency

Counts are given for total number of subjects, not for events

Counts are given by closest relationship (ie subjects experiencing more than 1

TEAE are counted only once within each SOC and PT using the most closely related event)

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: Similar table will be produced for Part 2 (ie Table 14.3.2.4)

Page x of y

TABLE 14.3.1.5
Subjects Reporting Adverse Drug Reactions
By MedDRA System Organ Class and Preferred Term
Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu$ g [14C]-KD025 IV infusion (N=X)

| - | | |
|-----------------------------|-----------|-------------|
| | n(%) | Events<br>n |
| Subjects Reporting ADRs (1) | xx (xx.x) | xx |
| SYSTEM ORGAN CLASS 1 | xx (xx.x) | xx |
| PREFFERED TERM 1 | xx (xx.x) | xx |
| PREFFERED TERM 2 | xx (xx.x) | xx |
| etc | | ••• |
| SYSTEM ORGAN CLASS 2 | xx (xx.x) | xx |
| PREFFERED TERM 1 | xx (xx.x) | xx |
| PREFFERED TERM 2 | xx (xx.x) | xx |
| etc | | *** |

Note: The data in this table are presented in listing x.x

- All subjects received a 200 mg KD025 oral tablet followed by 100 ug [14C]-KD025 IV infusion in Part 1
- (1) An ADR is any AE that the investigator considers possibly related or related to the IMP
- ADRs are coded using MedDRA v22.0 and are presented in descending order of frequency

Subjects experiencing more than 1 episode of an ADR are counted only once within each SOC and PT

Event is the total number of ADRs within the relevant SOC and PT

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: Counts of number of subjects are by maximum severity (ie using the most severe episode)
Programming note: Similar table will be produced for serious AEs and Part 2 (ie Table 14.3.1.6, 14.3.2.5 and 14.3.2.6)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.4.1.1 Haematology

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu$ g [14C]-KD025 IV Infusion (N=X)

<Parameter> (<units>) [ref range xxx - xxx (male)]

| | | _ | |
|----|------|-----|------|
| Dα | ~ ** | 7 | + |
| πe | | . Т | . L. |

#### Change from Baseline

| Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| BASELINE<br>Day 3 | xx | xx.xx<br>xx.xx | xx.xx<br>xx.xx | xx.xx<br>xx.xx | xx.x<br>xx.x | xx.x<br>xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 BASELINE is defined as Day 1, Pre-dose

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all haematology parameters and all time points.

Programming note: A similar table will be produced for Clinical Chemistry and Part 2 (ie Table 14.4.1.3, 14.4.2.1

and 14.4.2.3 - note that the post-baseline time point is different for Part 2, update table accordingly)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.4.1.2 Haematology

Shift Table: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu g$  [14C]-KD025 IV Infusion (N=X)

<Parameter> (<units>) [ref range xxx - xxx (male)]

#### Baseline

| Time Point<br>Assessment | n# | Below<br>n(%) | Within<br>n(%) | Above<br>n(%) |
|---|---|---|---|---|
| Day 3 | xx | | | |
| Below | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Within | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Above | | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 BASELINE is defined as Day 1, Pre-dose

N# is the total number of subjects that have a value at baseline and each given time-point and is used in the denominator for calculating the percentages of subjects, n indicates the number of subjects with a baseline and a post baseline assessment at the time point indicated. Below/within/above indicate the number (%) of subjects with assessments below/within/above the normal reference range

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all haematology parameters and all time points.

Programming note: A similar table will be produced for Clinical Chemistry and Part 2 (ie Table 14.4.1.4, 14.4.2.2 and 14.4.2.4 - note that the post-baseline time point is different for Part 2, update table accordingly)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.5.1.1 Vital Signs

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu$ g [14C]-KD025 IV Infusion (N=X)

<Parameter> (<units>) [ref range xxx - xxx (male)]

| | | | Char<br>Bas | Substantial<br>Change (1) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max | DEC | NONE | INC |
| BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | | | | |
| TIME POINT 1 | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx | xx |
| TIME POINT 2 | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx | xx |
| TIME POINT 3 | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx | xx |
| *** | *** | ••• | *** | ••• | ••• | ••• | | | ••• | ••• | ••• | | | | |
| <all other="" points="" time=""></all> | YY | YY YY | VV VV | VV VV | VV V | XX.X | vv | VV VV | ** ** | VV VV | VV V | vv v | vv | vv | vv |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 BASELINE is defined as Day 1, Pre-dose

(1) Substantial change is defined as: increase/decrease  $> \pm 20$  mmHg Systolic BP,  $> \pm 10$  mmHg Diastolic BP and  $> \pm 15$  bpm HR. DEC: number of subjects with substantial decrease from baseline NONE: number of subjects with no substantial change from baseline, INC: number of subjects with substantial increase from baseline

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Programming note: This table will be continued for all vital signs parameters and may be continued over more than one page Programming note: A similar table will be produced for Part 2 (ie Table 14.5.2.1)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.5.1.2.1

ECGs

Summary Statistics: Safety Population

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100 µg [14C]-KD025 IV Infusion (N=X)

<Parameter> (<units>) [ref range xxx - xxx (male)]

| Time Point | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| BASELINE | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | | | | | | |
| TIME POINT 1 | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x |
| TIME POINT 2 | XX | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x |
| TIME POINT 3 | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x |
| *** | | | | ••• | ••• | ••• | ••• | *** | ••• | *** | ••• | |
| <all other="" points="" time=""></all> | xx | xx.xx | XX.XX | xx.xx | xx.x | xx.x | xx | xx.xx | xx.xx | xx.xx | xx.x | xx.x |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 BASELINE is defined as Day 1, Pre-dose

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

DDMMMYYYY HH:MM

Change from Baseline

Programming note: This table will be continued for all ECG parameters and may be continued over more than one page

Programming note: Parameter may be added as the first column in this table.

Programming note: A similar table will be produced for Part 2 (ie Table 14.5.2.2.1)

Kadmon Corporation LLC Protocol: KD025-108

Page x of y

TABLE 14.5.1.2.2

ECGs

QTcF Categorical Data

Part 1: KD025 Oral Tablet & [14C]-KD025 IV Infusion

200 mg KD025 Oral Tablet & 100  $\mu$ g [14C]-KD025 IV Infusion (N=X)

<Parameter> (<units>) [ref range xxx - xxx (male)]

| | | | ~ | cF<br>.s (msec) | | | QTcF Interval<br>Increase (msec | |
|---|---|---|---|---|---|---|---|---|
| Time Point | N# | <=450<br>n(%) | 451-480<br>n(%) | 481-500<br>n(%) | >500<br>n(%) | <30<br>n(%) | 30-60<br>n(%) | >60<br>n(%) |
| BASELINE TIME POINT 1 TIME POINT 2 TIME POINT 3 | xx<br>xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| <all other="" points="" time=""></all> | <br>xx | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) |

Note: The data in this table are presented in listing x.x

All subjects received a 200 mg KD025 oral tablet followed by 100  $\mu$ g [14C]-KD025 IV infusion in Part 1 BASELINE is defined as Day 1, Pre-dose

Categories for QTcF interval and QTcF interval increases are based on ICH E14 guidelines

N# is the total number of subjects at the relevant time point and is used in the denominator for calculating the percentages of subjects, n indicates the number of subjects with observations at the given time point

PROGRAM PATH: X:\~\QSC200323\~\TFLS\PRODUCTION\TAB XX

Programming note: A similar table will be produced for Part 2 (ie Table 14.5.2.2.1)

# **Appendix 1: Part 1 Study Flow Chart**

| Study Day | S | Α | | | | | | | Res | sident ir | n Clinic | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| • | -28 to -2 | -1 | | | | | | | | 1 | | | | | | | , |
| Timepoint relative Oral Dosing (h) | | | P | 0 | 0.5 | 0.75 | 1 | 1.5 | 1.75 | 1.83 | 1.92 | 2 | 2.08 | 2.16 | 2.25 | 2.5 | 2.75 |
| Timepoint relative to end of IV infusion (h) | | | | | | | | | -0.25 | -0.16 | -0.08 | 0 | 0.08 | 0.16 | 0.25 | 0.5 | 0.75 |
| General Assessments | , | | | | | | | | * | 1 | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | |
| Medical History | X | Х | | | l | | | | | | | | | | <u> </u> | <u> </u> | <u> </u> |
| Weight and Height (including BMI) | X | | | | | | | | | | | | | | | | |
| Vein Assessment | X | | | | | | | | | | | | | | | | |
| CO Breath Test | Х | Х | | | | | | | | | | | | | | | <u> </u> |
| Drug Screen | X | X | | | | | | | | | | | | | | | |
| Alcohol Breath Test | Х | Х | | | | | | | | | | | | | | | |
| KD025 Oral Administration | | | | Х | | | | | | | | | | | | | |
| [ <sup>14</sup> C]-KD025 IV Administration | | | | | | | | | Xa | | | | | | | | |
| Safety Assessments | | | | | 2 - 2 2 | : | | | 3 - 2 - 1 | | | | | | | | |
| Physical Examination | X | | | | | | | | | | | | | | | | <u> </u> |
| Safety Labs <sup>b</sup> | X | | Х | | | | | | | | | | İ | | | | |
| Urinalysis | Х | | Х | | | | l | | | | | | | | | | |
| ECG | Х | Х | Х | | | | | | | | | | | | | | |
| Vital Signs <sup>c</sup> | Х | Х | Х | | | | | | | | | | <u> </u> | | <u> </u> | | |
| Adverse Events | - | | | | | | | | | | | | | | | | <u> </u> |
| Prior and Concomitant Medication | 4 | | | | | | | | | | | | | | | | <b>→</b> |
| PK and Total Radioactivity Assessments | | | | | | | | | | | | | | | | | |
| Plasma Samples for KD025 <sup>d</sup> | | | Х | | X | | Х | Х | | | | Х | | | | | |
| Plasma samples for [14C]-KD025e | | | | | | | | | Х | Х | Х | X | X | Х | X | Х | Х |

# Appendix 1 Part 1 Study Flow Chart (Continued)

| Study Day | | | | | | Re | side | nt in | Clinic | | | | | | D |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 1 | | | | | | | | 2 | 3 |
| Timepoint relative Oral Dosing (h) | 3 | 3.5 | 3.75 | 4 | 5 | 5.75 | 6 | 7 | 8 | 10 | 12 | 14 | 24 | 36 | 48 <sup>g</sup> |
| Timepoint relative to end of IV infusion (h) | 1 | 1.5 | 1.75 | 2 | 3 | 3.75 | 4 | 5 | 6 | 8 | 10 | 12 | 22 | 34 | <b>46</b> <sup>g</sup> |
| Safety Assessments | | | | | | | : | | | | | | | | |
| Physical Examination | | | ľ – | | | | | 1 | | | | | | | Xf |
| Safety Labs <sup>b</sup> | | | | | | | | <del>\ </del> | | | | | | | Х |
| Jrinalysis | | | | | | <u> </u> | | <del> </del> | | | | | | | Х |
| ECG | | | Х | | | X | - | <b></b> - | | | <b></b> | | Х | | Х |
| √ital Signs <sup>c</sup> | | | Х | | - | X | | <u> </u> | | | | | X | | Х |
| Adverse Events | 4 | <u> </u> | | | | <u> </u> | | | · | | <u> </u> | l | | IL | |
| Prior and Concomitant Medication | 4 | | | | | | | | | | | | | | |
| PK and Total Radioactivity Assessments | | | | . : | 1 | | | | | | | <u> </u> | ······································ | 1 | |
| Plasma Samples for KD025 <sup>d</sup> | X | <u> </u> | 1 | X | Х | | X | <u> </u> | Х | X | Х | | X | X | X |
| Plasma samples for [ <sup>14</sup> C]-KD025 <sup>e</sup> | X | X | | Х | х | | Х | Х | Х | Х | Х | Х | Х | Х | Х |

<sup>&</sup>lt;sup>14</sup>C: carbon-14, A: Admission, BMI: Body mass index, CO: carbon monoxide, D: Discharge, ECG: Electrocardiogram; IV: intravenous, P: pre-dose, S: Screening, 0.08 h: 5 min, 0.16 h: 10 min. Footnotes on next page

<sup>a</sup> 15 min IV infusion of [<sup>14</sup>C]-KD025 solution to be given 1.75 h post oral dose.

<sup>b</sup> Haematology and clinical chemistry at each time point including virology at screening. Creatinine clearance will be estimated at screening from serum creatinine using the Cockcroft-Gault equation.

Blood pressure, heart rate and oral temperature will be measured at the time points indicated above relative to the start of the infusion.

<sup>d</sup> All post-dose time points are relative to the oral KD025 dose

<sup>e</sup> All post-dose time points are relative to the end of the [<sup>14</sup>C]-KD025 infusion.

<sup>f</sup>Targeted (symptom driven) physical examination

<sup>9</sup> Discharge from clinical unit

## **Appendix 2: Part 2 Study Flow Chart**

| Study Day | Aª | | | | | | | | | R | esid | ent | in C | linic | | | | | | | | Dο | FUP° |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -1 | | | | | | | 1 | | | | | | | : | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 13-15 |
| | | Р | | | | | | | T | ime | Rel | ativ | e to | KD0 | 25 D | osing | (h) | | | | ··· | | |
| | | | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | 8 | 10 | 12 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | |
| General Assessments | <del></del> | - | | - <del></del> | | | | | | <u> </u> | | - | | | | _ | | 1 | | | <b></b> | | · |
| Medical History | Χ | | | | | | | | | Г | | | | | | | | | | | | | |
| Body Weight | X | | | | | | | | | | | | | | | | | | | | | | |
| CO Breath Test | X | | | | | | | | | | | | | | | | | | | | | | |
| Drug Screen | Х | | | | | | | | | | | | | | | | | | | | | | |
| Alcohol Breath Test | Х | | | | | | | | | | | | | | | | | | | | | | |
| [ <sup>14</sup> C]-KD025 Administration | | | X | | | | | | | | | | | | | | | | | | | | |
| Safety Assessments | | ; | | | | | | | | | | | | | | | | | | | | | <del></del> |
| Physical Examination <sup>d</sup> | ` | | | | | - | | <u> </u> | | | | | <u> </u> | | | | | | | | | X | <del></del> |
| Safety Labs <sup>e</sup> | | X | | | | | | | | | | | | | | | | | | | | Х | |
| Urinalysis | | X | Π | | | | | | | | | | | | | - | | | | | | Х | |
| ECG | X | X | | | | | Х | | Х | · | | | | | Х | | | | | | | X | |
| Vital Signs <sup>f</sup> | X | X | | | | | X | | Х | | | | | | Х | | | | | | | Х | |
| Adverse Events | | 4 | | | | | | | | | | | | | | | | | | | | | |
| Prior and Concomitant Medication | | 4 | | | | | | | | | | | | | | | | | | | | | <b>→</b> |
| Mass Balance and PK<br>Assessments | | | | | | | | | | | | | | | | | | | | | | | |
| Plasma Samples for KD025, KD025m1,<br>KD025m2 and TR | | х | | Х | х | Х | х | х | х | х | Х | X | х | Х | Х | Х | Х | Х | х | х | х | Х | |
| Whole blood samples for TR | | X | | | Х | | | | Х | | | Х | | Х | Х | | Х | Х | Х | Х | Х | Χ | |
| Plasma Samples for Metabolite Profiling and ID | | х | | | х | | | | х | | | Х | | Х | х | | Х | Х | х | х | х | Х | |
| Urine Samples for TR <sup>g</sup> | • | | | | | | | | | | | | | | | | | | | | <b>→</b> | | |
| Faecal Samples for TRh | | F | | | | | | _ | | _ | | | | | | | | | | | <b>→</b> | | |

<sup>&</sup>lt;sup>14</sup>C: carbon-14, A: Admission, CO: carbon monoxide, D: Discharge, ECG: Electrocardiogram, FUP: Follow-up visit/call, ID: Identification, P: Pre-dose, TR: total radioactivity. Footnotes on next page

<sup>a</sup> Subjects who participated in Part 1 will be admitted to the clinical unit after a minimum washout period of 7 days.

<sup>b</sup> Discharge from clinical unit. Subjects may be discharged as a group earlier if a cumulative mass balance recovery of >90% has been achieved or if <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 h periods. If the mass balance criteria have not been met by all subjects on Day 8, the residency period for the subjects not achieving the release criteria may be extended by up to a maximum of 2 additional 24 h periods (up to 216 h post-dose, Day 10) for further collection of urine and faeces. If the criteria are not met by Day 10, or if any additional residency is not considered appropriate or necessary, then home collections of urine and/or faeces may be requested at the discretion of the investigator for individual subjects.

<sup>c</sup> A follow-up phone call will take place 5 to 7 days after discharge or after the end of the last collection period.

<sup>d</sup> Targeted (symptom driven) physical examination

e Haematology and clinical chemistry at each time point.

f Blood pressure, heart rate and oral temperature will be measured at each time point

<sup>9</sup> A single urine sample will be collected at pre-dose (the first void of the day) and then during the following collection periods 0-6, 6-12, 12-24 h post-dose and then daily (24 h collections) until Day 8/Discharge.

h Faeces will be collected from admission until pre-dose and then daily (24 h collections) until Day 8/Discharge.